CLINICAL TRIAL: NCT00689936
Title: A Phase III, Randomized, Open-label, 3-arm Study to Determine the Efficacy and Safety of Lenalidomide(REVLIMID) Plus Low-dose Dexamethasone When Given Until Progressive Disease or for 18 Four-week Cycles Versus the Combination of Melphalan, Prednisone, and Thalidomide Given for 12 Six-week Cycles in Patients With Previously Untreated Multiple Myeloma Who Are Either 65 Years of Age or Older or Not Candidates for Stem Cell Transplantation.
Brief Title: Study to Determine Efficacy and Safety of Lenalidomide Plus Low-dose Dexamethasone Versus Melphalan, Prednisone, Thalidomide in Patients With Previously Untreated Multiple Myeloma
Acronym: FIRST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-020; 2007-004823-39 (EudraCT Number)
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed multiple myeloma; Lenalidomide; Revlimid; phase III
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone; Melphalan; Prednisone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lenalidomide / Dexamethasone until disease progression (Experimental): Lenalidomide plus low-dose dexamethasone given until disease progression
  Interventions: Drug: Lenalidomide and low-dose dexamethasone
- Lenalidomide / Dexamethasone for 18 cycles (Experimental): Lenalidomide plus low-dose dexamethasone given for 18 four-week cycles
  Interventions: Drug: Lenalidomide plus low-dose dexamethasone given for 18 four-week cycles
- Melphalan, Prednisone, and Thalidomide (MPT) for 12 cycles (Active Comparator): Combination of Melphalan, Prednisone and Thalidomide given for 12 six-week cycles
  Interventions: Drug: Melphalan, Prednisone and Thalidomide

INTERVENTIONS:
Drug: Lenalidomide and low-dose dexamethasone — Lenalidomide - oral, 2.5mg, 5mg, 10mg, 15mg 20mg, or 25 mg capsules, given either days 1-21 of each 28 day cycles or given every other day for 21 days until documentation of PD.
  Dexamethasone - oral 4mg tablets for a total dose of 20mg or 40 mg given days 1,8,15 and 22 of each 28 day cycle up to disease progression
  Other Names: Revlimid
  Arms: Lenalidomide / Dexamethasone until disease progression
Drug: Lenalidomide plus low-dose dexamethasone given for 18 four-week cycles — lenalidomide - oral, 2.5mg, 5mg, 10mg, 15mg, 20 mg or 25 mg capsules given on days 1-21 of each 28 day cycle or every other day for 21 days for 18 cycles.
  Dexamethasone - oral 4mg tablets for a total dose of 20mg or 40 mg given days 1,8,15 and 22 of each 28 day cycle for 18 cycles
  Other Names: Revlimid
  Arms: Lenalidomide / Dexamethasone for 18 cycles
Drug: Melphalan, Prednisone and Thalidomide — Melphalan - oral, 2mg tablets dosed at either 0.25mg/kg, 0.125 mg/kg, 0.20mg/kg or 0.10mg/kg on days 1-4 of each 42 day cycle up to 12 cycles Prednisone - oral, 5mg, 10mg, 20 mg and 50 mg tablets dosed at 2mg/kg daily days 1-4 of each 42 day cycle for up to 12 cycles Thalidomide - oral, 50mg, 100mg and 200 mg capsules dosed at either 100mg or 200 mg daily on days 1-41 of each 42 day cycle for up to 12 cycles
  Other Names: Prednisone; Thalomid
  Arms: Melphalan, Prednisone, and Thalidomide (MPT) for 12 cycles

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Lenalidomide plus low dose dexamethasone to that of the combination of melphalan, prednisone and thalidomide.

DETAILED DESCRIPTION:
CC-5013-MM020/IFM 07-01 is a Phase III, multicenter, randomized, open-label, 3-arm study that will compare the efficacy and safety of two Lenalidomide plus low-dose dexamethasone regimens given for two different durations of time (i.e., until progressive disease [PD] or for up to a maximum of 18 four-week cycles) to that of MPT given for a maximum of 12 six-week cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign informed consent form
2. Age ≥ 18 years at the time of signing consent
3. Previously untreated, symptomatic multiple myeloma as defined by the 3 criteria below:

   * MM diagnostic criteria (all 3 required):
   * Monoclonal plasma cells in the bone marrow ≥10% and/or presence of a biopsy-proven plasmacytoma
   * Monoclonal protein present in the serum and/or urine
   * Myeloma-related organ dysfunction (at least one of the following) [C] Calcium elevation in the blood (serum calcium >10.5 mg/dl or upper limit of normal) [R] Renal insufficiency (serum creatinine >2 mg/dl) [A] Anemia (hemoglobin <10 g/dl or 2 g < laboratory normal) [B] Lytic bone lesions or osteoporosis

   AND have measurable disease by protein electrophoresis analyses as defined by the following:
   * IgG multiple myeloma: Serum monoclonal paraprotein (M-protein) level ≥ 1.0 g/dl or urine M-protein level ≥ 200 mg/24 hours
   * IgA multiple myeloma: Serum M-protein level ≥ 0.5 g/dl or urine M-protein level ≥ 200 mg/24 hours
   * IgM multiple myeloma (IgM M-protein plus lytic bone disease documented by skeletal survey plain films): Serum M-protein level ≥ 1.0 g/dl or urine M-protein level ≥ 200mg/24hours
   * IgD multiple myeloma: Serum M-protein level ≥ 0.05 g/dl or urine M-protein level ≥ 200 mg/24 hours
   * Light chain multiple myeloma: Serum M-protein level ≥ 1.0 g/dl or urine M-protein level ≥ 200 mg/24 hours

   AND are at least 65 years of age or older or, if younger than 65 years of age, are not candidates for stem cell transplantation because:
   * The patient declines to undergo stem cell transplantation or
   * Stem cell transplantation is not available to the patient due to cost or other reasons
4. ECOG performance status of 0, 1, or 2
5. Able to adhere to the study visit schedule and other protocol requirements
6. Females of child-bearing potential (FCBP)^2:

   1. Must agree to undergo two medically supervised pregnancy tests prior to starting study therapy with either Rd or MPT. The first pregnancy test will be performed within 10-14 days prior to the start of Rd or MPT and the second pregnancy test will be performed within 24 hours prior to the start of Rd or MPT. She must also agree to ongoing pregnancy testing during the course of the study and after the end of study therapy. This applies even if the patient practices complete and continued sexual abstinence.
   2. Must commit to either continued abstinence from heterosexual intercourse (which must be reviewed on a monthly basis) or agree to use and be able to comply with effective contraception without interruption, 28 days prior to starting study drug, during the study therapy (including during periods of dose interruptions), and for 28 days after discontinuation of study therapy.
7. Male Patients:

   1. Must agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after cessation of study therapy.
   2. Must agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
   3. Must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
8. All patients must:

   1. Have an understanding that the study drug could have a potential teratogenic risk.
   2. Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy.
   3. Agree not to share study medication with another person. All FCBP and male patients must be counseled about pregnancy precautions and risks of fetal exposure.

Exclusion Criteria:

1. Previous treatment with anti-myeloma therapy (does not include radiotherapy, bisphosphonates, or a single short course of steroid [i.e., less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days; such a short course of steroid treatment must not have been given within 14 days of randomization]).
2. Any serious medical condition that places the patient at an unacceptable risk if he or she participates in this study. Examples of such a medical condition are, but are not limited to, patient with unstable cardiac disease as defined by: Cardiac events such as MI within the past 6 months, NYHA heart failure class III-IV, uncontrolled atrial fibrillation or hypertension; patients with conditions requiring chronic steroid or immunosuppressive treatment, such as rheumatoid arthritis, multiple sclerosis and lupus, that likely need additional steroid or immunosuppressive treatments in addition to the study treatment.
3. Pregnant or lactating females.
4. Any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,000/µL (1.0 x 109/L)
   * Untransfused platelet count < 50,000 cells/µL (50 x 10^9/L)
   * Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)
5. Renal failure requiring hemodialysis or peritoneal dialysis.
6. Prior history of malignancies, other than multiple myeloma, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

   * Basal cell carcinoma of the skin
   * Squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
7. Patients who are unable or unwilling to undergo antithrombotic therapy.
8. Peripheral neuropathy of > grade 2 severity.
9. Known HIV positivity or active infectious hepatitis, type A, B, or C. Primary AL (immunoglobulin light chain) amyloidosis and myeloma complicated by amyloidosis.

   * 1 A variety of other types of end organ dysfunctions can occasionally occur and lead to a need for therapy. Such dysfunction is sufficient to support classification as myeloma if proven to be myeloma-related.
   * 2 A FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (i.e., amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1623 (Actual)
Dates: Start 2008-08-21 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2016-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jacques, MD, Study Director — Celgene Corporation
Locations (288):
- United States (32):
  - University of AL Birmingham, Birmingham, Alabama
  - Cedar Sinai Medical Center Dept of Medicine, Los Angeles, California
  - University of California, San Francisco- California, San Francisco, California
  - Stanford University Stanford, Stanford, California
  - Gainesville Heme Oncology Associates, Gainesville, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Integrated Community Oncology Network, Orange Park, Florida
  - Gulf Coast Oncology, St. Petersburg, Florida
  - Palm Beach Cancer Institute, LLC, West Palm Beach, Florida
  - Southern Illinois Hematology Oncology, Centralia, Illinois
  - Orchard Healthcare Research, Inc., Chicago, Illinois
  - John H Stroger Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Ingalls Cancer Institute, Harvey, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Maine Center for Cancer Medicine Blood Disorders, Scarborough, Maine
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Billings Clinic, Billings, Montana
  - Arena Oncology Associates, PC, Lake Success, New York
  - Dakota Cancer Institute, Fargo, North Dakota
  - Gabrail Cancer Center Research, Canton, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Kaiser Permanente Northwest Oncology Hematology, Portland, Oregon
  - St. Luke's Hospital and Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Cancer Center, Collierville, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (17):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre Divsion of Haematology Medical Oncology, East Melbourne, Victoria
  - Western Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Flinders Medical Centre, Bedford Park
  - Geelong Hospital, Geelong
  - Gosford Hospital, Gosford
  - Royal Brisbane and Women's Hospital, Herston
  - Cabrini Hospital, Malvern
  - The Royal Melbourne Hospital, Parkville
  - Royal Perth Hospital, Perth
  - Gold Coast Hospital, Southport
  - Royal North Shore Hospital, St Leonards
  - Westmead Hospital, Wentworthville
  - Border Medical Oncology, Wodonga
  - Wollongong Hospital, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Austria (11):
  - Hospital Leoben, Leoben
  - Hospital of Barmherzige Schwestern Linz, Linz
  - Hospital of Elisabethinen Linz, Linz
  - General Hospital Linz, Linz
  - MM-015. Salzburger Landkliniken, St. Johanns-Spital, Universitätsklinik fur Innere Medizin III, Salzburg
  - Hospital St. Polten, Sankt Pölten
  - Hospital of the Barmherzigen Bruder Vienna, Vienna
  - MM-015.Wihelminenspital, Vienna
  - MM-015. Medizinische Universität Wien, Vienna
  - Hospital Wels, Wels
  - Hospital Wiener Neustadt, Wiener Neustadt
- Belgium (13):
  - ZNA Stuivenberg Centrumziekenhuis, Antwerp
  - Les Cliniques du Sud Luxembourg, Arlon
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Jules Bordet Institut, Brussels
  - Hopital Erasme, Brussels
  - AZ-VUB, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
  - Virga Jesse Ziekenhuis, Hasselt
  - Universitair Ziekenhuis Leuven, Campus Gasthuisberg, Leuven
  - H. Hartziekenhuis Roeselare-Menen vzw campus Wilgenstraat, Roeselare
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Canada (23):
  - University of Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Kelowna, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - BC Cancer Agency - Fraser Valley Centre, Surrey, British Columbia
  - Leukemia/BMT Program of BCDiv of Hem, Vancouver Gen Hosp, Vancouver, British Columbia
  - Vancouver Island Cancer Center, Victoria, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Science Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hospital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - Hotel-Dieu de Levis, Lévis, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Hospital Maisonneuve - Rosemont, Montreal, Quebec
  - CHUM- Hopital Notre-Dame, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Sir Mortimer B. Davis - Jewish Genl, Montreal, Quebec
  - CHUQ - Hotel-Dieu de QuebecHematology - Oncology, Québec
- China (5):
  - Chaoyang Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Ruijin Hospital Shanghai Jiaotong University, Shanghai
  - Blood Disease Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Tianjin
- France (68):
  - Clinique Claude BernardOncologie, Albi
  - CHU Sud, Amiens
  - CHRU Hopital du bocage, Angers
  - CH Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier de la cote basque, Bayonne
  - Centre Hospitalier, Blois
  - Hopital Avicenne, Bobigny
  - Institut Bergonie Centre Regional de Lutte Contre Le Cancer de Bordeaux Et Sud Ouest, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital de Fleyriat, Bourg-en-Bresse
  - Hopital Augustin Morvan, Brest
  - CHU, Caen
  - Centre Francois Baclesse, Caen
  - CH, Cannes
  - CH Rene Dubois, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon/Saone Cedex
  - Hopital Antoine Beclere, Clamart
  - Hopital dinstruction des armees Percy, Clamart
  - Chu Estaing, Clermont-Ferrand
  - CH Louis Pasteur, Colmar
  - Hopital Henri Mondor, Créteil
  - CHRU Hopital du bocage, Dijon
  - Centre Hospitalier General, Dunkirk
  - Institut Prive de Cancerologie, Grenoble
  - CHRU, Grenoble
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - CH, Le Chesnay
  - Hopital J MonodRhumato Nord, Le Havre
  - Kremlin Bicetre, Le Kremlin-Bicêtre
  - Centre Jean Bernard, Le Mans
  - Centre Hospitalier, Le Mans
  - GH de Institut Catholique St Vincent, Lille
  - CHRU-Hopital Claude Huriez, Lille
  - CH - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - CHU Hopital Edouard Herriot, Lyon
  - Centre Hospitalier de Valence, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hopital de Mercy, Metz
  - Clinique Pont de chaume Oncologie et Radiotherapie, Montauban
  - CHU Montpellier - Hôpital Lapeyronie, Montpellier
  - Hopital Emile Muller, Mulhouse
  - CHRU - Hotel Dieu, Nantes
  - Centre Antoine Lacassagne Oncologie medicale et Hematologie, Nice
  - Hopital de lArchet 1, Nice
  - CH La Source, Orléans
  - Hopital Saint Louis, Paris
  - Hopital Necker, Paris
  - CHU Hôpital St-Antoine, Paris
  - Hopital Cochin, Paris
  - CHRU - Hopital du Haut Leveque, Pessac
  - CU CHU Clemenceau, Poitiers
  - Hopital R. Debre, Reims
  - CHU Reims - Hôpital Maison Blanche, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - CHRU Hopital sud Medecine Interne, Rennes
  - CHG Rodez, Rodez
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de Loire, Saint-Priest-en-Jarez
  - CHRU Hôpital de Hautepierre, Strasbourg
  - CHRU Hopital Purpan, Toulouse
  - CHRU Hopital Bretonneau, Tours
  - CHRU Hopital Trousseau, Tours
  - CHRU Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CH P. Chubert, Vannes
  - Institut Gustave Roussy, Villejuif
- Germany (17):
  - Medizinische Kinik und Poliklinik I, Dresden
  - Universitaetsklinikum Dusseldorf Klinik fuer Haematologie, Düsseldorf
  - Universitatsklinikum Essen-, Essen
  - Staedtische Kliniken Frankfurt am Main Hochst, Frankfurt am Main
  - Universitatsklinikum Giessen, Giessen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Askepios Klinik St. Georg, Hamburg
  - Universitatsklinikum Jena, Jena
  - Medizinische Klinik und Poliklinik II, Leipzig
  - Universitatsklinikum schleswig-Holstein, Lübeck
  - Klinikum der Johann-Wolfgang-Goethe-Universtat, München
  - Medizinische Klinik III Klinikum der Universität München-Großhadern, München
  - Poliklinik A, Münster
  - Medizinische Fakultat der Universitat Rostock, Rostock
  - Zentrum F. Innere Medizin II Robert- Bosch-Krankenhaus GmBH, Stuttgart
  - Medizinische Klinik - Abteilung II, Tübingen
  - Klinik fur Innere Medizin III, Ulm
- Greece (6):
  - Alexandra Hospital, University of Athens, Athens
  - Attiko Hospital of Athens, Athens
  - Evangelismos Hospital of Athens, Athens
  - University of Athens, Athens
  - Metaxa Hospital Peiraias, Piraeus
  - Theagenio Anticancer Hospital of Thessaloniki, Thessaloniki
- Ireland (3):
  - Adelaide and Meath Hospital, Dublin
  - Mater Misercordiae Hospital, Dublin
  - University Hospital Galway, Galway
- Italy (18):
  - Policlinico S. Orsola, Bologna
  - Oncologia Medica, Università della Magna Grecia, Catanzaro
  - Clinica Ematologica, A.O.U. San Martino di Genova, Genova
  - Ematologia ed Immunologia, Azienda Ospedaliera Vito Fazzi di Lecce, Lecce
  - Unità Operativa di Oncoematologia, Ospedale di Matera, Matera
  - U.O. di Ematologia e Trapianto di Midollo Osseo, Milan
  - Istituto Europeo di Oncologia - IEO, Milan
  - Presidio Ospedaliero A. Perrino, Milan
  - Policlinico di Modena, Modena
  - Oncoematologia, Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Casa di Cura La Maddalena, Divisione di Ematologia, Palermo
  - Policlinico San Matteo Universita Di Pavia, Pavia
  - Ospedale Civile, Piacenza
  - A.O. Universitaria Ospedale S.Chiara Dip.Oncologia, Div. Ematologia, Pisa
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Istituto Nazionale Tumori Regina Elena, Struttura Complessa Ematologia ed Unita di Cellule Staminali, Roma
  - Azienda Policlinico Umberto I, Universita La Sapienzadi Roma, Rome
  - Ospedale Molinette, Torino
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Newtown
- Portugal (6):
  - Hospital de Sao Marcos, Braga
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Instituto Português de Oncologia Porto, Porto
  - Hospital de Santo Antonio- Porto, Porto
- South Korea (15):
  - Hallym University Sacred Heart Hospital, Anyang
  - Inje University Busan Paik Hospital, Busan
  - Daegu Catholic University Medical Center 3056-6, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Gyeonggi-do
  - Hwasun Chonnam National University Hospital, Hwasun-goon
  - Gachon University Gil Hospital, Incheon
  - Chonbuk National University Hospital 42, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Seongsanno
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul - Saint Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (20):
  - Hospital Universitari Germans Trias i Pujol, Badalona (Barcelona)
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Instituto Catalan de Oncologia-Hospital Duran, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital de Donosti, Donostia / San Sebastian
  - Hospital Univ. Josep Trueta, Girona
  - Hospital Clinico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Messeguer, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Clinica Universitaria de Navarra,, Pamplona
  - Hospital Sant Pau, Reus
  - Hospital Universtario Marques de Valdecilla, Santander
  - Hospital Clinico Santiago de Compostela, Santiago de Compostela
  - Hosptial La Fe, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- Sweden (4):
  - Linkoping University Hospital, Linköping
  - Karolinska University HospitalSolna, Stockholm
  - St. Görans Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
- Switzerland (7):
  - Abteilung Onkologie Haematologie des Kantonsspitals Aarau, Aarau
  - UniversitatsSpital Basel, Basel
  - Inselsspital Bern, Bern
  - Kantonsspital Graubunden, Chur
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital Munsterlingen, Münsterlingen
  - Kantonsspital Winterthur, Winterthur
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Veteran General Hospital - Taipei, Taipei
  - National Taiwan University Hospital, Tapei
- United Kingdom (17):
  - Gwynedd Hospital, Bangor
  - Royal United Hospital, Bath
  - Belfast City Hospital Haematology Department, Belfast Northern Ireland
  - Birminghman QE, Birmingham West Midlands
  - Royal Bournemouth Hosp, Bournemouth Dorset
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales - Cardiff, Cardiff
  - The Beatson West of Scotland Centre, Glasgow
  - Dept of Haematology St Bartholomews Hospital, London
  - Guy's and St Thomas' Hospital - London, London
  - Royal Free Hospital, London
  - Churchhill Hospital, Oxford
  - Derriford Hospital, Plymouth Crownhill Devon
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Trust, Sheffield
  - Pinderfields General Hospital, West Yorkshire
  - New Cross Hospital- Wolverhampton, Wolverhampton

REFERENCES:
- [Background] Dimopoulos MA, Cheung MC, Roussel M, Liu T, Gamberi B, Kolb B, Derigs HG, Eom H, Belhadj K, Lenain P, Van der Jagt R, Rigaudeau S, Dib M, Hall R, Jardel H, Jaccard A, Tosikyan A, Karlin L, Bensinger W, Schots R, Leupin N, Chen G, Marek J, Ervin-Haynes A, Facon T. Impact of renal impairment on outcomes with lenalidomide and dexamethasone treatment in the FIRST trial, a randomized, open-label phase 3 trial in transplant-ineligible patients with multiple myeloma. Haematologica. 2016 Mar;101(3):363-70. doi: 10.3324/haematol.2015.133629. Epub 2015 Dec 11. PMID 26659916
- [Background] Hulin C, Belch A, Shustik C, Petrucci MT, Duhrsen U, Lu J, Song K, Rodon P, Pegourie B, Garderet L, Hunter H, Azais I, Eek R, Gisslinger H, Macro M, Dakhil S, Goncalves C, LeBlanc R, Romeril K, Royer B, Doyen C, Leleu X, Offner F, Leupin N, Houck V, Chen G, Ervin-Haynes A, Dimopoulos MA, Facon T. Updated Outcomes and Impact of Age With Lenalidomide and Low-Dose Dexamethasone or Melphalan, Prednisone, and Thalidomide in the Randomized, Phase III FIRST Trial. J Clin Oncol. 2016 Oct 20;34(30):3609-3617. doi: 10.1200/JCO.2016.66.7295. PMID 27325857
- [Background] Delforge M, Minuk L, Eisenmann JC, Arnulf B, Canepa L, Fragasso A, Leyvraz S, Langer C, Ezaydi Y, Vogl DT, Giraldo-Castellano P, Yoon SS, Zarnitsky C, Escoffre-Barbe M, Lemieux B, Song K, Bahlis NJ, Guo S, Monzini MS, Ervin-Haynes A, Houck V, Facon T. Health-related quality-of-life in patients with newly diagnosed multiple myeloma in the FIRST trial: lenalidomide plus low-dose dexamethasone versus melphalan, prednisone, thalidomide. Haematologica. 2015 Jun;100(6):826-33. doi: 10.3324/haematol.2014.120121. Epub 2015 Mar 13. PMID 25769541
- [Background] Benboubker L, Dimopoulos MA, Dispenzieri A, Catalano J, Belch AR, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis N, Banos A, Tiab M, Delforge M, Cavenagh J, Geraldes C, Lee JJ, Chen C, Oriol A, de la Rubia J, Qiu L, White DJ, Binder D, Anderson K, Fermand JP, Moreau P, Attal M, Knight R, Chen G, Van Oostendorp J, Jacques C, Ervin-Haynes A, Avet-Loiseau H, Hulin C, Facon T; FIRST Trial Team. Lenalidomide and dexamethasone in transplant-ineligible patients with myeloma. N Engl J Med. 2014 Sep 4;371(10):906-17. doi: 10.1056/NEJMoa1402551. PMID 25184863
- [Background] Vogl DT, Delforge M, Song K, Guo S, Gibson CJ, Ervin-Haynes A, Facon T. Long-term health-related quality of life in transplant-ineligible patients with newly diagnosed multiple myeloma receiving lenalidomide and dexamethasone. Leuk Lymphoma. 2018 Feb;59(2):398-405. doi: 10.1080/10428194.2017.1334125. Epub 2017 Jun 22. PMID 28641472
- [Background] Dumontet C, Hulin C, Dimopoulos MA, Belch A, Dispenzieri A, Ludwig H, Rodon P, Van Droogenbroeck J, Qiu L, Cavo M, Van de Velde A, Lahuerta JJ, Allangba O, Lee JH, Boyle E, Perrot A, Moreau P, Manier S, Attal M, Roussel M, Mohty M, Mary JY, Civet A, Costa B, Tinel A, Gaston-Mathe Y, Facon T. A predictive model for risk of early grade >/= 3 infection in patients with multiple myeloma not eligible for transplant: analysis of the FIRST trial. Leukemia. 2018 Jun;32(6):1404-1413. doi: 10.1038/s41375-018-0133-x. Epub 2018 Apr 26. PMID 29784907
- [Background] Ailawadhi S, Jacobus S, Sexton R, Stewart AK, Dispenzieri A, Hussein MA, Zonder JA, Crowley J, Hoering A, Barlogie B, Orlowski RZ, Rajkumar SV. Disease and outcome disparities in multiple myeloma: exploring the role of race/ethnicity in the Cooperative Group clinical trials. Blood Cancer J. 2018 Jul 6;8(7):67. doi: 10.1038/s41408-018-0102-7. PMID 29980678
- [Background] Jain T, Sonbol MB, Firwana B, Kolla KR, Almader-Douglas D, Palmer J, Fonseca R. High-Dose Chemotherapy with Early Autologous Stem Cell Transplantation Compared to Standard Dose Chemotherapy or Delayed Transplantation in Patients with Newly Diagnosed Multiple Myeloma: A Systematic Review and Meta-Analysis. Biol Blood Marrow Transplant. 2019 Feb;25(2):239-247. doi: 10.1016/j.bbmt.2018.09.021. Epub 2018 Sep 20. PMID 30244101
- [Background] Facon T, Dimopoulos MA, Dispenzieri A, Catalano JV, Belch A, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis NJ, Banos A, Tiab M, Delforge M, Cavenagh JD, Geraldes C, Lee JJ, Chen C, Oriol A, De La Rubia J, White D, Binder D, Lu J, Anderson KC, Moreau P, Attal M, Perrot A, Arnulf B, Qiu L, Roussel M, Boyle E, Manier S, Mohty M, Avet-Loiseau H, Leleu X, Ervin-Haynes A, Chen G, Houck V, Benboubker L, Hulin C. Final analysis of survival outcomes in the phase 3 FIRST trial of up-front treatment for multiple myeloma. Blood. 2018 Jan 18;131(3):301-310. doi: 10.1182/blood-2017-07-795047. Epub 2017 Nov 17. PMID 29150421
- [Background] Ailawadhi S, DerSarkissian M, Duh MS, Lafeuille MH, Posner G, Ralston S, Zagadailov E, Ba-Mancini A, Rifkin R. Cost Offsets in the Treatment Journeys of Patients With Relapsed/Refractory Multiple Myeloma. Clin Ther. 2019 Mar;41(3):477-493.e7. doi: 10.1016/j.clinthera.2019.01.009. Epub 2019 Feb 14. PMID 30773308
- [Background] Pegourie B, Karlin L, Benboubker L, Orsini-Piocelle F, Tiab M, Auger-Quittet S, Rodon P, Royer B, Leleu X, Bareau B, Cliquennois M, Fuzibet JG, Voog E, Belhadj-Merzoug K, Decaux O, Rey P, Slama B, Leyronnas C, Zarnitsky C, Boyle E, Bosson JL, Pernod G; IFM Group. Apixaban for the prevention of thromboembolism in immunomodulatory-treated myeloma patients: Myelaxat, a phase 2 pilot study. Am J Hematol. 2019 Jun;94(6):635-640. doi: 10.1002/ajh.25459. Epub 2019 Apr 1. PMID 30859608
- [Result] Bahlis NJ, Corso A, Mugge LO, Shen ZX, Desjardins P, Stoppa AM, Decaux O, de Revel T, Granell M, Marit G, Nahi H, Demuynck H, Huang SY, Basu S, Guthrie TH, Ervin-Haynes A, Marek J, Chen G, Facon T. Benefit of continuous treatment for responders with newly diagnosed multiple myeloma in the randomized FIRST trial. Leukemia. 2017 Nov;31(11):2435-2442. doi: 10.1038/leu.2017.111. Epub 2017 Apr 4. PMID 28373701
- [Result] Lu J, Lee JH, Huang SY, Qiu L, Lee JJ, Liu T, Yoon SS, Kim K, Shen ZX, Eom HS, Chen WM, Min CK, Kim HJ, Lee JO, Kwak JY, Yiu W, Chen G, Ervin-Haynes A, Hulin C, Facon T. Continuous treatment with lenalidomide and low-dose dexamethasone in transplant-ineligible patients with newly diagnosed multiple myeloma in Asia: subanalysis of the FIRST trial. Br J Haematol. 2017 Mar;176(5):743-749. doi: 10.1111/bjh.14465. Epub 2017 Jan 20. PMID 28106903
- See also: Link to CSR synopsis — http://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/clinical-study-report-csr-synopses/purposes-of-posting-clinical-study-report-csr-synopses

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the Europe, Asia, North America and Pacific regions. Participants were randomized at 246 sites (165 in Europe, 23 in Asia, 39 in North America, and 19 in the Pacific). The study was co-sponsored by Intergroupe Francophone du Myélome (IFM) (for sites in France, Switzerland, and Belgium) and Celgene Corporation.
Pre-assignment Details: Participants were stratified at randomization by 1) age (≤ 75 versus > 75 years), 2) stage (International Staging System Stages I or II versus Stage III), and 3) country.
Groups:
- Lenalidomide and Low-Dose Dexamethasone (Rd): Participants ≤ 75 years old received 25 mg lenalidomide (R) administered by mouth (PO) on days 1 to 21 of each 28-day cycle plus 40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle until disease progression or intolerable toxicity. Participants > 75 years old received lenalidomide 25 mg PO on the same schedule and frequency plus 20 mg dexamethasone at the same schedule. Participants with moderate renal insufficiency received 10-15 mg lenalidomide (R) PO on days 1-21 of each 28-day treatment cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle until disease progression or intolerable toxicity. Participants with severe renal insufficiency received 15 mg lenalidomide (R) PO every other day on days 1-21 of each 28-day treatment cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle until disease progression or intolerable toxicity.
- Lenalidomide and Dexamethasone Rd18: Participants ≤ 75 years old received 25 mg lenalidomide (R) PO on days 1 to 21 of each 28-day treatment cycle 40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless progressive disease (PD) or intolerable toxicity occurred. Those > 75 years old received lenalidomide 25 mg PO on the same schedule and frequency plus 20 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity. Those with moderate renal insufficiency received 10-15 mg lenalidomide (R) PO on days 1-21 of each 28-day cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity. Participants with severe renal insufficiency received 15 mg lenalidomide (R) PO every other day (QOD) on days 1-21 of each 28-day cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity.
- Melphalan + Prednisone + Thalidomide (MPT): Participants received melphalan (M) 0.25 mg/kg PO daily (QD) on days 1 to 4 of each 42-day cycle plus prednisone (P) at 2 mg/kg PO on days 1 to 4 of each 42-day cycle and thalidomide 200 mg PO QD on days 1 to 41 of each 42-day cycle. MPT therapy was given for up to 12 cycles unless PD or intolerable toxicity occurred. Participants with moderate to severe renal insufficiency received melphalan (M) 0.10-0.125 mg/kg PO daily (QD) on days 1 to 4 of each 42-day cycle plus prednisone (P) at 2 mg/kg PO on days 1 to 4 of each 42-day cycle and thalidomide 100-200 mg PO QD on days 1 to 41 of each 42-day cycle. MPT therapy was given for up to 12 cycles unless PD or intolerable toxicity occurred.
Period: Active Treatment Phase
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Started | 535 | 541 | 547
Safety Population | 532 (Safety population = all randomized participants who received at least 1 dose of study treatment.) | 540 (Safety population = all randomized participants who received at least 1 dose of study treatment.) | 541 (Safety population = all randomized participants who received at least 1 dose of study treatment.)
Untreated | 3 (Participants randomized, but did not receive any study drug treatment.) | 1 (Participants randomized, but did not receive any study drug treatment.) | 6 (Participants randomized, but did not receive any study drug treatment.)
Completed | 0 | 0 | 0
Not Completed | 535 | 541 | 547
Not completed — Adverse Event | 68 | 71 | 76
Not completed — Disease Progression | 273 | 362 | 339
Not completed — Withdrawal by Subject | 16 | 16 | 21
Not completed — Death | 60 | 28 | 37
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Protocol Violation | 2 | 2 | 4
Not completed — Study Close Out | 64 | 26 | 21
Not completed — Miscellaneous | 52 | 34 | 47
Period: Progression Free Survival-PFS-Follow-Up
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Started | 87 (Includes participants who discontinued treatment for reasons other than progressive disease.) | 300 (Includes participants who completed 18 cycles (Rd18) and did not experience progressive disease.) | 273 (Includes participants who completed 12 cycles MPT and did not experience progressive disease.)
Completed | 87 | 300 | 273
Not Completed | 0 | 0 | 0
Period: Long-Term Follow Up Phase
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Started | 382 (Includes participants from both the active treatment phase and from the PFS follow-up phase.) | 463 (Includes participants from both the active treatment phase and from the PFS follow-up phase.) | 459 (Includes participants from both the active treatment phase and from the PFS follow-up phase.)
Completed | 255 | 275 | 315
Not Completed | 127 | 188 | 144
Not completed — Continue in Long Term Follow Up | 127 | 188 | 144

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population includes all participants who were randomized, independent of whether they received study treatment or not
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT) | Total
Number analyzed (Participants) | 535 | 541 | 547 | 1623
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (6.57) | 72.9 (6.50) | 73.1 (6.32) | 73.1 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 268 | 260 | 769
  Male | 294 | 273 | 287 | 854
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 40 | 43 | 44 | 127
  Black or African American | 9 | 6 | 5 | 20
  Native Hawaiian or other Pacific Islanders | 1 | 0 | 1 | 2
  White or Caucasian | 474 | 480 | 491 | 1445
  Other, Miscellaneous | 6 | 11 | 3 | 20
  Undisclosed | 5 | 1 | 3 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 37 | 33 | 36 | 106
  Not Hispanic or Latino | 493 | 505 | 508 | 1506
  Undisclosed | 5 | 3 | 3 | 11
International Staging System (ISS) [Number; unit: Participants] — International Staging System (ISS) is used as a staging system for multiple myeloma and divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels. Higher stages represent more advanced disease.
  Participants
    Stage I | 106 | 106 | 103 | 315
    Stage II | 227 | 229 | 225 | 681
    Stage III | 202 | 206 | 219 | 627
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used to assess the progress of disease in a patient, how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  Participants
    0 (fully active) | 155 | 163 | 156 | 474
    1 (restrictive but ambulatory) | 257 | 263 | 275 | 795
    2 (ambulatory but unable to work) | 119 | 113 | 111 | 343
    3-4 (limited self-care, completely disabled) | 2 | 2 | 2 | 6
    Missing | 2 | 0 | 3 | 5
Creatinine clearance [Number; unit: Participants]
  >=60 ml/min | 269 | 280 | 285 | 834
  <60 ml/min | 266 | 261 | 261 | 788
  Missing | 0 | 0 | 1 | 1
Beta2 Microglobulin [Number; unit: Participants]
  >5.5 mg/L | 224 | 224 | 234 | 682
  <=5.5 mg/L | 309 | 316 | 312 | 937
  Missing | 2 | 1 | 1 | 4
Albumin [Number; unit: Participants]
  <=35 g/L | 192 | 209 | 223 | 624
  > 35 g/L | 343 | 331 | 324 | 998
  Missing | 0 | 1 | 0 | 1
Lactic Dehydrogenase [Number; unit: Participants]
  <200 U/L | 448 | 442 | 434 | 1324
  >=200 U/L | 86 | 99 | 112 | 297
  Missing | 1 | 0 | 1 | 2
Multiple Myeloma Subtype [Number; unit: Participants]
  Immunoglobulin A | 138 | 142 | 123 | 403
  Immunoglobulin A and Immunoglobulin G | 7 | 6 | 8 | 21
  Immunoglobulin A and Immunoglobulin M | 0 | 0 | 1 | 1
  Immunoglobulin D | 4 | 7 | 4 | 15
  Immunoglobulin G | 334 | 331 | 350 | 1015
  Immunoglobulin M | 3 | 1 | 1 | 5
  Not available (includes light-chain disease) | 49 | 54 | 60 | 163
Cytogenetic Risk [Number; unit: Participants] — Cytogenetic risk categories are mutually exclusive. Definitions: Adverse risk category: t(4:14), t(14:16), del (13q) or monosomy 13, del (17p), 1q gain; Non-adverse risk categories include favorable hyperdiploidy: t(11:14), gains of 5/9/15; normal: a normal result, gains other than 5/9/15, IgH deletion, and uncertain risk: probes used for analysis cannot place participant in any risk categories. Not evaluable: no specimen received, test failure or insufficient number of cells available for analysis.
  Participants
    Adverse Risk | 170 | 185 | 189 | 544
    Favorable Hyperdiploidy | 112 | 103 | 102 | 317
    Normal | 148 | 131 | 141 | 420
    Uncertain Risk | 38 | 56 | 40 | 134
    Not evaluable | 34 | 35 | 44 | 113
    Missing | 33 | 31 | 31 | 95

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates of Progression-free Survival (PFS) Based on the Response Assessment by the Independent Review Adjudication Committee (IRAC)
Description: PFS was calculated as the time from randomization to the first documented PD or death due to any cause during the study, which ever occurred first based on the International Myeloma Working Group Uniform Response criteria (IMWG). Those who withdrew for any reason or received another anti-myeloma therapy without documented PD were censored on the date of their last response assessment, prior to receiving any other anti-myeloma therapy. Censoring rules for PFS: - No baseline assessments and no progression or death documented within the 2 scheduled assessments; Death within the lst two assessments without any adequate response assessment; Progression documented between scheduled assessments; Death between adequate assessments; no progression; study discontinuations for reasons other than PD or death; new anti-myeloma started prior to PD; death or PD after an extended lost to follow-up time period (2 or more missed scheduled assessment's).
Time Frame: From date of randomization until the data cut-off date of 24 May 2013. Median follow-up time for all participants was 17.1 months.
Population: The intent to treat (ITT) population included all participants who were randomized, independent of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 25.5 [20.7 to 29.4] | 20.7 [19.4 to 22.0] | 21.2 [19.3 to 23.2]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00006, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.61 to 0.85] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.60 to 0.82] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.70349, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.89 to 1.20] — Based on stratified Cox proportional hazards model comparing the hazard functions associated with treatment groups

2. Primary Outcome: Kaplan-Meier Estimates of PFS Based on the Response Assessment by the Investigator At the Time of Final Analysis
Description: as for outcome 1
Time Frame: From date of randomization to date of data cut-off date of 21 January 2016; median follow-up for all participants was 17.7 months
Population: The intent to treat population included all participants who were randomized, independent of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 26.0 [20.7 to 29.7] | 21.0 [19.7 to 22.4] | 21.9 [19.8 to 23.9]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.59 to 0.79] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.60 to 0.81] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.91161, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.14] — Based on a stratified Cox proportional hazards model

3. Secondary Outcome: Kaplan Meier Estimates of Overall Survival at the Time of Final Analysis (OS)
Description: Overall survival was defined as the time between randomization and death. Participants, who died, regardless of the cause of death, were considered to have had an event. All participants who were lost to follow-up prior to the end of the trial or who were withdrawn from the trial were censored at the time of last contact. Participants who were still being treated were censored at the last available date the participant was known to be alive.
Time Frame: From date of randomization to date of data cut-off date of 21 January 2016; median follow-up for all participants was 48.3 months
Population: ITT population included all participants who were randomized, independent of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 59.1 [53.9 to 65.9] | 62.3 [53.6 to 68.7] | 49.1 [44.3 to 53.5]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00234, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.67 to 0.92] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.82903, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.86 to 1.20] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00119, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.66 to 0.90] — Based on a stratified Cox proportional hazards model

4. Secondary Outcome: Percentage of Participants With an Objective Response Based on IRAC Review
Description: Objective response according to IMWG Uniform Response Criteria was defined as a best overall response including a complete response (CR), very good partial response (VGPR) or partial response (PR) based on the IRAC Review. A CR is defined as: negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in BM; A VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; A PR is: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. If present at baseline a ≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: Disease response was assessed every 28 days until end of treatment or the data cut-off date of 24 May 2013; median duration of treatment was 80.2 weeks in the Rd arm; 72 weeks in the Rd18 arm and 67.1 weeks in the MPT arm
Population: ITT population includes all participants who were randomized, independent of whether they received study treatment or not.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
percentage of participants | 75.1 | 73.4 | 62.3
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Fisher Exact; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.41 to 2.37]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.53065, Fisher Exact; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.83 to 1.44]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00010, Fisher Exact; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.29 to 2.15]

5. Secondary Outcome: Percentage of Participants With an Objective Response Based on Investigator Assessment at Time of Final Analysis
Description: Objective response according to IMWG Uniform Response Criteria was defined as a best overall response including a complete response (CR), very good partial response (VGPR) or partial response (PR) based on the IRAC Review. A CR is defined s: negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in BM; A VGPR is serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; A PR is: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. If present at baseline a ≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: Disease response was assessed every 28 days until end of treatment or the data cut-off date of 21 January 2016; median duration of treatment was 80.2 weeks in the Rd arm; 72 weeks in the Rd18 arm and 67.1 weeks in the MPT arm
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
percentage of participants | 80.7 | 78.6 | 67.5
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Fisher Exact; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.53 to 2.68]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.40500, Fisher Exact; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.85 to 1.54]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00004, Fisher Exact; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.35 to 2.32]

6. Secondary Outcome: Kaplan Meier Estimates of Duration of Myeloma Response as Determined by the IRAC
Description: Duration of response was defined as the duration from the time when the response criteria were first met for CR or VGPR or PR based on IMWG criteria until the first date the response criteria were met for progressive disease or until the participant died from any cause, whichever occurred first.
Time Frame: Disease response was assessed every 28 days until end of treatment or the data cut-off date of 24 May 2013; median follow-up for responders was 20.1 months
Population: Study participants with at least a PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 402 | 397 | 341
months | 35.0 [27.9 to 43.4] | 22.1 [20.3 to 24.0] | 22.3 [20.2 to 24.9]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.51 to 0.76] — Based on unstratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.50 to 0.72] — Based on unstratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.76740, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.86 to 1.23] — Based on unstratified Cox proportional hazards model

7. Secondary Outcome: Kaplan Meier Estimates of Duration of Myeloma Response as Determined by an Investigator Assessment at Time of Final Analysis
Description: as for outcome 6
Time Frame: Disease response was assessed every 28 days until end of treatment; data cut-off date of 21 January 2016; median follow-up for responders was 19.9 months
Population: Study participants with at least a PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 432 | 425 | 369
months | 31.5 [26.2 to 37.3] | 21.5 [19.2 to 23.0] | 22.1 [20.3 to 24.5]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.51 to 0.72] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.52 to 0.72] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.99537, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.85 to 1.17] — Based on a stratified Cox proportional hazards model

8. Secondary Outcome: Time to First Response Based on the Review by the IRAC
Description: The time to first myeloma response was defined as the time from randomization to the time when the response criteria for at least a PR was first met based on the IMWG criteria.
Time Frame: as for outcome 4
Population: Participants who had at least a PR.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 402 | 397 | 341
months | 1.8 [0.7 to 22.2] | 1.8 [0.8 to 17.1] | 2.8 [1.3 to 49.7]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.46672, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Time to First Response Based on the Investigator Assessment at the Time of Final Analysis
Description: The time to first myeloma response was defined as the time from randomization to the time when the response criteria for at least a PR was first met based on the IMWG criteria assessed by the investigator.
Time Frame: as for outcome 5
Population: Participants who had at least a PR.
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 430 | 425 | 368
months | 1.8 [0.5 to 22.2] | 1.8 [0.8 to 34.8] | 2.8 [1.2 to 56.3]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.46987, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Kaplan Meier Estimates of Time to Treatment Failure (TTF)
Description: TTF is defined as the time between the randomization and discontinuation of study treatment for any reason, including disease progression (determined by IRAC based on the IMWG response criteria), treatment toxicity, start of another anti-myeloma therapy (AMT) or death.
Time Frame: From date of randomization until the data cut-off of 24 May 2013; median follow-up for all participants was 16.1 months.
Population: ITT population includes participants who were randomized, independent of whether they received study treatment or not
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 16.9 [14.1 to 18.4] | 17.2 [14.6 to 18.2] | 14.1 [12.0 to 16.1]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00012, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.68 to 0.88] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.00187, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.71 to 0.93] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.45973, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.84 to 1.08] — Based on a stratified Cox proportional hazards model

11. Secondary Outcome: Kaplan Meier Estimates of Time to Treatment Failure (TTF) at the Time of Final Analysis
Description: TTF is defined as the time between the randomization and discontinuation of study treatment for any reason, including disease progression (determined by the investigators assessment based on the IMWG response criteria), treatment toxicity, start of another anti-myeloma therapy (AMT) or death.
Time Frame: From date of randomization until the data cut-off date of 21 January 2016; median follow up for all participants was 16.1 months.
Population: ITT population includes participants who were randomized, independent of whether they received study treatment or not
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 16.9 [14.1 to 18.4] | 17.2 [14.6 to 18.2] | 14.1 [12.0 to 16.1]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00002, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.67 to 0.86] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.00126, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.72 to 0.92] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.27704, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.83 to 1.06] — Based on a stratified Cox proportional hazards model

12. Secondary Outcome: Kaplan Meier Estimates for Time to Second-line Anti-myeloma Treatment (AMT)
Description: Time to second-line anti-myeloma therapy was defined as time from randomization to the start of another non-protocol anti-myeloma therapy.
Time Frame: From date of randomization until the data cut-off of 24 May 2013; median follow-up for all participants was 23.0 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 39.1 [32.8 to NA] — Could not be estimated due to the low number of events at the time of analysis | 28.5 [26.9 to 30.4] | 26.7 [24.0 to 29.9]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.56 to 0.78] — Based on a stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.00067, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.88] — Based on a stratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.12333, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.75 to 1.03] — Based on a stratified Cox proportional hazards model

13. Secondary Outcome: Kaplan Meier Estimates of Time to Second Line Therapy AMT at the Time of Final Analysis
Description: Time to second-line anti-myeloma therapy is defined as time from randomization to the start of another non-protocol anti-myeloma therapy. Those who do not receive another anti-myeloma therapy were censored at the last assessment or follow-up visit known to have received no new therapy.
Time Frame: From date of randomization until the data cut-off of date 21 January 2016; median follow-up for all participants was 23.0 months
Population: as for outcome 4
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 535 | 541 | 547
months | 36.7 [31.9 to 45.2] | 28.5 [26.9 to 30.4] | 26.7 [24.0 to 29.1]
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p < 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.54 to .73] — Based on unstratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.00001, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.61 to 0.83] — Based on unstratified Cox proportional hazards model
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.05821, Log Rank — The p-value is based on the unstratified log-rank test; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.76 to 1.00] — Based on unstratified Cox proportional hazards model

14. Secondary Outcome: Percentage of Participants With an Objective Response After Second-line Anti-myeloma Treatment at the Time of Final Analysis
Description: as for outcome 5
Time Frame: Disease response was assessed every 28 days until end of treatment; data cut-off date of 21 January 2016; median duration of treatment was 80.2 weeks in the Rd arm; 72 weeks in the Rd18 arm and 67.1 weeks in the MPT arm
Population: ITT population; Participants with second line AMT.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 299 | 377 | 381
percentage of participants | 46.2 | 53.1 | 45.7
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.93824, Fisher Exact; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.75 to 1.38]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.08836, Fisher Exact; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.56 to 1.03]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.04974, Fisher Exact; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.01 to 1.79]

15. Secondary Outcome: Percentage of Participants With a Myeloma Response by Adverse Risk Cytogenetic Risk Category Based on IRAC Review.
Description: Participants were placed in adverse and non-adverse cytogenetic risk categories at baseline and response rates evaluated. Adverse Risk: t(4;14), t(14;16), del(13q) or monosomy 13, del(17p), 1q gain Favorable Hyperdiploidy: : t(11;14), gains of 5/9/15; Normal: a normal result, gains other than 5/9/15, IgH deletion Uncertain risk: probes used for analysis cannot place participant in any of the other risk categories. Objective response = best overall response including CR, VGPR or PR based on the IRAC Review; A CR is negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in BM; A VGPRis serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; A PR is ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. If present at baseline a ≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: as for outcome 4
Population: ITT population with Cytogenetic risk of Adverse Risk
Measure: Number; unit: Percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 170 | 185 | 189
Percentage of participants | 70.0 | 69.7 | 58.2
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.02134, Fisher Exact; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.08 to 2.59]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 1.00000, Fisher Exact; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.64 to 1.59]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.02374, Fisher Exact; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.08 to 2.53]

16. Secondary Outcome: Percentage of Participants With a Myeloma Response by Favorable Hyperdiploidy Risk Cytogenetic Risk Category Based on IRAC Review
Description: as for outcome 15
Time Frame: as for outcome 4
Population: ITT population with a Cytogenetic Risk of Favorable Hyperploidy
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 112 | 103 | 102
percentage of participants | 80.4 | 81.6 | 70.6
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.11152, Fisher Exact; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.91 to 3.21]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.86336, Fisher Exact; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.47 to 1.83]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.07321, Fisher Exact; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.96 to 3.55]

17. Secondary Outcome: Percentage of Participants With a Myeloma Response by Normal Risk Cytogenetic Risk Category Based on IRAC Review
Description: as for outcome 15
Time Frame: as for outcome 4
Population: ITT population with a cytogenetic risk of normal
Measure: Number; unit: percentage of particpants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 148 | 131 | 141
percentage of particpants | 80.4 | 74.8 | 61.0
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.00043, Fisher Exact; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.55 to 4.45]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.31274, Fisher Exact; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.78 to 2.43]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.01936, Fisher Exact; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.13 to 3.19]

18. Secondary Outcome: Percentage of Participants With a Myeloma Response by Uncertain Risk Cytogenetic Risk Category Based on IRAC Review
Description: as for outcome 15
Time Frame: as for outcome 4
Population: ITT population with a Cytogenetic Risk of Uncertain Risk
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 38 | 56 | 40
percentage of participants | 60.5 | 76.8 | 57.5
Statistical Analysis 1: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.82128, Fisher Exact; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.46 to 2.80]
Statistical Analysis 2: Comparison: Lenalidomide and Low-Dose Dexamethasone (Rd) vs Lenalidomide and Dexamethasone Rd18; Test type: Superiority or Other; p = 0.11041, Fisher Exact; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.19 to 1.14]
Statistical Analysis 3: Comparison: Lenalidomide and Dexamethasone Rd18 vs Melphalan + Prednisone + Thalidomide (MPT); Test type: Superiority or Other; p = 0.07302, Fisher Exact; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.01 to 5.91]

19. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Health Status Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status/QOL scale is scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in QOL or functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 508 | 507 | 508
units on a scale
  Month 1: number analyzed (Participants) | 438 | 441 | 415
  Month 1 | 0.4 (23.98) | -1.3 (23.93) | 1.0 (23.68)
  Month 3: number analyzed (Participants) | 421 | 413 | 396
  Month 3 | 4.8 (24.15) | 4.7 (25.15) | 4.3 (26.04)
  Month 6: number analyzed (Participants) | 369 | 376 | 351
  Month 6 | 5.9 (25.93) | 5.4 (23.88) | 6.1 (25.98)
  Month 12: number analyzed (Participants) | 302 | 299 | 252
  Month 12 | 4.8 (26.42) | 3.2 (25.38) | 6.5 (25.90)
  Month 18: number analyzed (Participants) | 246 | 238 | 178
  Month 18 | 6.4 (28.02) | 5.7 (24.86) | 4.8 (27.05)
  Study discontinuation: number analyzed (Participants) | 203 | 261 | 257
  Study discontinuation | -0.1 (27.07) | 5.0 (27.33) | 0.3 (28.07)

20. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Physical Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 511 | 514 | 509
units on a scale
  Month 1: number analyzed (Participants) | 445 | 449 | 419
  Month 1 | -1.7 (21.11) | -1.4 (19.56) | -0.9 (21.28)
  Month 3: number analyzed (Participants) | 426 | 421 | 396
  Month 3 | 3.4 (23.33) | 4.7 (22.94) | 2.2 (23.68)
  Month 6: number analyzed (Participants) | 376 | 382 | 352
  Month 6 | 4.7 (25.09) | 7.6 (22.85) | 5.3 (24.52)
  Month 12: number analyzed (Participants) | 307 | 302 | 253
  Month 12 | 5.0 (25.65) | 7.4 (23.40) | 6.9 (27.22)
  Month 18: number analyzed (Participants) | 247 | 243 | 183
  Month 18 | 6.9 (26.71) | 6.8 (23.58) | 8.3 (27.10)
  Discontinuation Visit: number analyzed (Participants) | 207 | 267 | 256
  Discontinuation Visit | -0.1 (29.70) | 3.0 (27.32) | -0.1 (27.58)

21. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Role Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Role Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 508 | 508
units on a scale
  Month 1: number analyzed (Participants) | 442 | 445 | 415
  Month 1 | -2.7 (29.94) | -4.6 (28.20) | -2.4 (30.48)
  Month 3: number analyzed (Participants) | 422 | 419 | 395
  Month 3 | 2.4 (33.32) | 6.3 (32.43) | 4.1 (34.23)
  Month 6: number analyzed (Participants) | 373 | 378 | 352
  Month 6 | 6.3 (35.44) | 8.6 (32.42) | 8.2 (36.09)
  Month 12: number analyzed (Participants) | 305 | 300 | 252
  Month 12 | 7.8 (36.60) | 9.4 (34.15) | 11.8 (38.94)
  Month 18: number analyzed (Participants) | 245 | 240 | 182
  Month 18 | 8.0 (35.34) | 9.1 (34.35) | 14.5 (39.03)
  Discontinuation Visit: number analyzed (Participants) | 206 | 264 | 256
  Discontinuation Visit | -0.3 (39.58) | 3.8 (36.34) | -1.0 (38.41)

22. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Emotional Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Emotional Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 510 | 510
units on a scale
  Month 1: number analyzed (Participants) | 443 | 446 | 419
  Month 1 | 0.6 (22.13) | 0.1 (20.73) | 1.0 (21.52)
  Month 3: number analyzed (Participants) | 423 | 415 | 397
  Month 3 | 3.8 (22.29) | 3.9 (22.11) | 2.1 (22.27)
  Month 6: number analyzed (Participants) | 375 | 379 | 351
  Month 6 | 4.6 (24.36) | 5.8 (22.39) | 5.5 (22.55)
  Month 12: number analyzed (Participants) | 305 | 301 | 254
  Month 12 | 4.6 (24.08) | 4.9 (22.23) | 5.1 (22.37)
  Month 18: number analyzed (Participants) | 246 | 242 | 179
  Month 18 | 5.8 (25.61) | 3.1 (23.31) | 5.1 (22.99)
  Discontinuation Visit: number analyzed (Participants) | 205 | 263 | 256
  Discontinuation Visit | 2.6 (24.30) | 3.7 (23.77) | -0.0 (24.72)

23. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Cognitive Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Cognitive Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1, (Baseline) then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 510 | 510
units on a scale
  Month 1: number analyzed (Participants) | 443 | 447 | 419
  Month 1 | -1.2 (21.73) | -1.7 (19.08) | -1.8 (24.07)
  Month 3: number analyzed (Participants) | 424 | 415 | 397
  Month 3 | -0.7 (22.89) | 1.8 (20.94) | -1.5 (24.02)
  Month 6: number analyzed (Participants) | 375 | 379 | 353
  Month 6 | -0.9 (22.57) | 0.9 (19.77) | -0.3 (23.55)
  Month 12: number analyzed (Participants) | 306 | 301 | 254
  Month 12 | -1.6 (25.05) | -1.2 (20.19) | -0.6 (22.97)
  Month 18: number analyzed (Participants) | 246 | 242 | 179
  Month 18 | -2.2 (25.61) | -2.8 (20.97) | -0.7 (23.99)
  Discontinuation Visit: number analyzed (Participants) | 206 | 263 | 256
  Discontinuation Visit | -4.9 (27.57) | -2.6 (22.34) | -7.1 (25.15)

24. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Social Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Social Functioning Scale is scored between 0 and 100, with a high score indicating better functioning/support. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 505 | 503 | 503
units on a scale
  Month 1: number analyzed (Participants) | 439 | 441 | 414
  Month 1 | -4.3 (29.10) | -2.2 (27.44) | -1.4 (30.52)
  Month 3: number analyzed (Participants) | 419 | 410 | 389
  Month 3 | 0.7 (29.36) | 2.0 (30.93) | 2.4 (30.70)
  Month 6: number analyzed (Participants) | 374 | 374 | 348
  Month 6 | 4.0 (32.48) | 5.2 (28.50) | 3.4 (35.24)
  Month 12: number analyzed (Participants) | 305 | 298 | 252
  Month 12 | 2.9 (34.96) | 3.8 (32.29) | 5.8 (33.68)
  Month 18: number analyzed (Participants) | 247 | 239 | 177
  Month 18 | 4.2 (34.99) | 3.2 (31.67) | 6.0 (35.20)
  Discontinuation Visit: number analyzed (Participants) | 204 | 257 | 254
  Discontinuation Visit | -1.2 (33.50) | 2.7 (33.37) | -3.5 (33.20)

25. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Fatigue Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate improvement in symptoms and positive values indicate worsening symptoms.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 511 | 514 | 512
units on a scale
  Month 1: number analyzed (Participants) | 445 | 448 | 421
  Month 1 | 2.6 (25.32) | 4.4 (24.03) | 2.8 (25.44)
  Month 3: number analyzed (Participants) | 425 | 423 | 400
  Month 3 | -2.5 (28.15) | -3.4 (25.16) | -1.8 (28.53)
  Month 6: number analyzed (Participants) | 376 | 383 | 355
  Month 6 | -3.7 (28.54) | -5.9 (26.37) | -4.5 (29.09)
  Month 12: number analyzed (Participants) | 306 | 303 | 255
  Month 12 | -4.3 (29.47) | -2.3 (26.63) | -3.9 (29.56)
  Month 18: number analyzed (Participants) | 244 | 242 | 184
  Month 18 | -3.1 (29.82) | 0.1 (29.12) | -4.3 (30.05)
  Discontinuation Visit: number analyzed (Participants) | 207 | 267 | 258
  Discontinuation Visit | 0.3 (29.75) | -1.6 (29.11) | 2.7 (30.15)

26. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Pain Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Pain Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate improvement in symptoms and positive values indicate worsening symptoms.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 511 | 514 | 512
units on a scale
  Month 1: number analyzed (Participants) | 446 | 453 | 423
  Month 1 | -5.4 (31.89) | -4.4 (30.70) | -7.8 (30.93)
  Month 3: number analyzed (Participants) | 426 | 423 | 399
  Month 3 | -13.4 (34.28) | -13.1 (32.32) | -12.1 (31.98)
  Month 6: number analyzed (Participants) | 379 | 384 | 355
  Month 6 | -14.4 (35.64) | -16.1 (33.44) | -13.4 (34.45)
  Month 12: number analyzed (Participants) | 306 | 304 | 255
  Month 12 | -14.0 (36.05) | -14.7 (32.34) | -14.3 (32.85)
  Month 18: number analyzed (Participants) | 248 | 242 | 183
  Month 18 | -14.4 (35.03) | -12.4 (35.28) | -14.7 (32.81)
  Discontinuation Visit: number analyzed (Participants) | 207 | 266 | 259
  Discontinuation Visit | -8.0 (39.37) | -7.9 (37.65) | -6.0 (37.09)

27. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Nausea/Vomiting Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Nausea/Vomiting Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate improvement in symptoms and positive values indicate worsening symptoms.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 511 | 513 | 512
units on a scale
  Month 1: number analyzed (Participants) | 446 | 449 | 424
  Month 1 | 1.8 (20.05) | -0.5 (23.19) | 4.0 (22.91)
  Month 3: number analyzed (Participants) | 426 | 422 | 399
  Month 3 | -1.1 (19.42) | -2.5 (21.92) | -1.2 (19.89)
  Month 6: number analyzed (Participants) | 377 | 381 | 355
  Month 6 | -1.3 (18.53) | -4.0 (21.52) | -3.9 (19.57)
  Month 12: number analyzed (Participants) | 306 | 302 | 255
  Month 12 | -2.2 (17.16) | -3.6 (18.86) | -3.9 (19.09)
  Month 18: number analyzed (Participants) | 246 | 242 | 184
  Month 18 | -2.3 (19.20) | -2.7 (18.92) | -3.9 (19.44)
  Discontinuation Visit: number analyzed (Participants) | 206 | 267 | 258
  Discontinuation Visit | 0.4 (21.43) | -4.2 (24.37) | 1.0 (21.46)

28. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Dyspnea Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnoea Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate improvement in symptoms and positive values indicate worsening symptoms.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population includes all participants with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 508 | 506
units on a scale
  Month 1: number analyzed (Participants) | 439 | 440 | 417
  Month 1 | 0.9 (30.87) | 3.6 (29.85) | 4.2 (32.04)
  Month 3: number analyzed (Participants) | 423 | 417 | 390
  Month 3 | -0.8 (31.87) | -1.9 (29.45) | 2.0 (32.49)
  Month 6: number analyzed (Participants) | 372 | 375 | 351
  Month 6 | -2.3 (33.12) | -2.9 (29.66) | 0.1 (30.29)
  Month 12: number analyzed (Participants) | 303 | 294 | 253
  Month 12 | -3.5 (30.97) | -1.6 (29.23) | -1.6 (32.76)
  Month 18: number analyzed (Participants) | 244 | 238 | 182
  Month 18 | -1.8 (32.73) | 2.9 (28.33) | 0.4 (32.68)
  Discontinuation Visit: number analyzed (Participants) | 204 | 262 | 255
  Discontinuation Visit | -1.0 (37.42) | 0.8 (31.01) | 7.8 (33.72)

29. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Insomnia Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Insomnia Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate improvement in symptoms and positive values indicate worsening symptoms.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: Intent to Treat (ITT) population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 510 | 513 | 511
units on a scale
  Month 1: number analyzed (Participants) | 443 | 447 | 421
  Month 1 | 2.1 (33.34) | 3.2 (34.32) | -10.5 (30.47)
  Month 3: number analyzed (Participants) | 422 | 420 | 399
  Month 3 | 0.2 (35.11) | -1.3 (33.54) | -8.9 (35.28)
  Month 6: number analyzed (Participants) | 379 | 382 | 353
  Month 6 | -1.2 (34.84) | -1.9 (31.43) | -11.6 (32.96)
  Month 12: number analyzed (Participants) | 303 | 300 | 253
  Month 12 | -1.0 (34.78) | 1.1 (32.47) | -9.6 (31.00)
  Month 18: number analyzed (Participants) | 243 | 241 | 182
  Month 18 | -0.5 (37.11) | 1.4 (35.72) | -6.0 (34.42)
  Discontinuation Visit: number analyzed (Participants) | 204 | 265 | 254
  Discontinuation Visit | -5.2 (36.47) | -1.6 (31.27) | -4.5 (36.98)

30. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Appetite Loss Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Appetite Loss Scale is scored between 0 and 100, with a high score indicating a higher level of appetite loss. Negative change from Baseline values indicate improvement in appetite and positive values indicate worsening of appetite.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 512 | 510
units on a scale
  Month 1: number analyzed (Participants) | 442 | 447 | 422
  Month 1 | 1.3 (33.46) | 2.9 (31.87) | 1.0 (32.35)
  Month 3: number analyzed (Participants) | 424 | 421 | 396
  Month 3 | -5.9 (38.34) | -3.3 (35.25) | -6.2 (35.03)
  Month 6: number analyzed (Participants) | 374 | 381 | 354
  Month 6 | -9.8 (40.02) | -8.6 (33.98) | -13.5 (35.98)
  Month 12: number analyzed (Participants) | 307 | 299 | 253
  Month 12 | -7.3 (37.07) | -6.4 (35.30) | -10.5 (34.16)
  Month 18: number analyzed (Participants) | 246 | 241 | 183
  Month 18 | -8.1 (35.97) | -5.1 (33.29) | -12.2 (31.88)
  Discontinuation Visit: number analyzed (Participants) | 203 | 267 | 257
  Discontinuation Visit | -1.0 (36.77) | -7.5 (37.49) | -2.6 (37.18)

31. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Constipation Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Constipation Scale is scored between 0 and 100, with a high score indicating a higher level of constipation. Negative change from Baseline values indicate improvement in constipation and positive values indicate worsening of constipation.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 508 | 511 | 510
units on a scale
  Month 1: number analyzed (Participants) | 441 | 446 | 419
  Month 1 | 8.3 (36.74) | 6.3 (36.18) | 18.4 (41.23)
  Month 3: number analyzed (Participants) | 422 | 416 | 397
  Month 3 | 1.8 (37.53) | 0.0 (37.02) | 13.9 (39.30)
  Month 6: number analyzed (Participants) | 373 | 377 | 353
  Month 6 | -2.4 (37.51) | -5.1 (37.39) | 6.8 (40.41)
  Month 12: number analyzed (Participants) | 304 | 301 | 255
  Month 12 | -2.4 (38.79) | -5.2 (38.09) | 3.7 (38.28)
  Month 18: number analyzed (Participants) | 246 | 242 | 179
  Month 18 | -4.5 (35.42) | -5.9 (36.65) | 0.0 (37.06)
  Discontinuation Visit: number analyzed (Participants) | 203 | 261 | 257
  Discontinuation Visit | -7.9 (39.98) | -7.5 (39.20) | -2.2 (38.86)

32. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Diarrhea Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Diarrhea Scale is scored between 0 and 100, with a high score indicating a higher level of diarrhea. Negative change from Baseline values indicate improvement in diarrhea and positive values indicate worsening of diarrhea.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 508 | 509 | 510
units on a scale
  Month 1: number analyzed (Participants) | 438 | 444 | 416
  Month 1 | 3.8 (25.53) | 2.3 (24.94) | -0.6 (18.79)
  Month 3: number analyzed (Participants) | 419 | 413 | 395
  Month 3 | 3.7 (24.99) | 3.4 (27.27) | -2.4 (18.61)
  Month 6: number analyzed (Participants) | 373 | 376 | 351
  Month 6 | 8.2 (28.36) | 6.0 (27.95) | -2.2 (21.19)
  Month 12: number analyzed (Participants) | 303 | 299 | 253
  Month 12 | 11.8 (31.35) | 9.1 (28.74) | -2.5 (17.26)
  Month 18: number analyzed (Participants) | 246 | 241 | 178
  Month 18 | 14.8 (31.20) | 10.9 (30.96) | -1.7 (17.46)
  Discontinuation Visit: number analyzed (Participants) | 206 | 261 | 255
  Discontinuation Visit | 10.8 (29.56) | 6.4 (31.38) | -0.5 (19.39)

33. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Financial Difficulties Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used in clinical research to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Financial Difficulties Scale is scored between 0 and 100, with a high score indicating a higher level of financial difficulties. Negative change from Baseline values indicate improvement in financial difficulties and positive values indicate worsening of financial difficulties.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 501 | 504 | 502
units on a scale
  Month 1: number analyzed (Participants) | 435 | 441 | 409
  Month 1 | 2.1 (21.43) | -0.3 (20.59) | 0.5 (22.98)
  Month 3: number analyzed (Participants) | 413 | 407 | 388
  Month 3 | 1.9 (23.09) | -0.4 (21.88) | 1.9 (21.48)
  Month 6: number analyzed (Participants) | 370 | 373 | 345
  Month 6 | 1.4 (22.92) | -0.3 (21.24) | 0.7 (24.57)
  Month 12: number analyzed (Participants) | 302 | 299 | 249
  Month 12 | 0.4 (23.99) | 1.6 (23.28) | 1.1 (23.16)
  Month 18: number analyzed (Participants) | 244 | 239 | 174
  Month 18 | 2.0 (22.23) | 1.8 (23.30) | 0.4 (21.20)
  Discontinuation Visit: number analyzed (Participants) | 197 | 255 | 254
  Discontinuation Visit | 1.9 (27.19) | 0.5 (23.84) | 5.0 (24.82)

34. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Disease Symptoms Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores were averaged, and transformed to a 0-100 scale; a higher score indicates more severe disease symptom(s).
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 510 | 512 | 511
units on a scale
  Month 1: number analyzed (Participants) | 442 | 448 | 421
  Month 1 | -4.0 (18.75) | -4.1 (19.37) | -4.4 (19.04)
  Month 3: number analyzed (Participants) | 422 | 418 | 396
  Month 3 | -9.1 (21.66) | -10.0 (19.97) | -7.0 (20.43)
  Month 6: number analyzed (Participants) | 375 | 381 | 353
  Month 6 | -8.8 (20.89) | -9.9 (20.94) | -7.9 (21.94)
  Month 12: number analyzed (Participants) | 306 | 303 | 254
  Month 12 | -7.8 (21.74) | -8.7 (20.29) | -6.5 (21.58)
  Month 18: number analyzed (Participants) | 249 | 243 | 183
  Month 18 | -8.7 (23.50) | -6.2 (23.30) | -7.9 (21.26)
  Discontinuation Visit: number analyzed (Participants) | 205 | 266 | 259
  Discontinuation Visit | -3.5 (24.82) | -4.5 (24.90) | -3.7 (23.54)

35. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Side Effects Treatment Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores were averaged, and transformed to a 0-100 scale; a higher score represents a more severe overall side effect of treatment.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 509 | 511 | 510
units on a scale
  Month 1: number analyzed (Participants) | 438 | 446 | 418
  Month 1 | 2.5 (13.72) | 4.0 (14.89) | 5.6 (15.00)
  Month 3: number analyzed (Participants) | 421 | 417 | 393
  Month 3 | 1.0 (15.23) | 1.2 (14.67) | 3.5 (15.40)
  Month 6: number analyzed (Participants) | 374 | 378 | 351
  Month 6 | 1.7 (15.58) | -0.4 (14.39) | 2.9 (17.28)
  Month 12: number analyzed (Participants) | 305 | 301 | 254
  Month 12 | 1.9 (14.49) | 1.2 (16.20) | 4.7 (17.17)
  Month 18: number analyzed (Participants) | 247 | 243 | 182
  Month 18 | 2.2 (15.63) | 2.3 (17.36) | 4.3 (16.37)
  Discontinuation Visit: number analyzed (Participants) | 205 | 262 | 258
  Discontinuation Visit | 0.6 (15.85) | -1.0 (15.81) | 3.8 (16.52)

36. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Future Perspective Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores were averaged, and transformed to a 0-100 scale; for the future perspective scale, a higher score indicates a better perspective of the future.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 504 | 508 | 509
units on a scale
  Month 1: number analyzed (Participants) | 433 | 443 | 415
  Month 1 | 4.7 (22.17) | 3.9 (20.94) | 3.3 (23.20)
  Month 3: number analyzed (Participants) | 416 | 414 | 394
  Month 3 | 8.5 (23.28) | 9.2 (22.95) | 6.3 (25.06)
  Month 6: number analyzed (Participants) | 367 | 377 | 350
  Month 6 | 9.8 (23.67) | 12.3 (24.84) | 8.0 (25.26)
  Month 12: number analyzed (Participants) | 303 | 299 | 249
  Month 12 | 10.8 (21.90) | 12.1 (24.41) | 10.0 (26.30)
  Month 18: number analyzed (Participants) | 245 | 239 | 179
  Month 18 | 12.7 (23.96) | 11.7 (24.76) | 9.5 (21.75)
  Discontinuation Visit: number analyzed (Participants) | 203 | 264 | 254
  Discontinuation Visit | 5.8 (25.91) | 8.8 (26.71) | 3.2 (27.13)

37. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Body Image Scale
Description: EORTC QLQ-MY20 is a validated questionnaire to assess the overall quality of life in patients with multiple myeloma. EORTC QLQ-MY20 includes four scales: disease symptoms, treatment side-effects, future perspective, and body image. Questions used a 4-point scale (from 1 'Not at All' to 4 'Very Much'). Scores were averaged, and transformed to a 0-100 scale; for the body image scale, a higher score indicates a better body image.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 492 | 498 | 504
units on a scale
  Month 1: number analyzed (Participants) | 417 | 422 | 408
  Month 1 | -4.5 (29.44) | -1.5 (27.19) | -1.6 (29.97)
  Month 3: number analyzed (Participants) | 404 | 398 | 387
  Month 3 | -1.7 (27.54) | 0.8 (26.23) | -3.0 (29.38)
  Month 6: number analyzed (Participants) | 357 | 366 | 347
  Month 6 | -1.4 (27.84) | 1.5 (29.72) | -2.8 (33.07)
  Month 12: number analyzed (Participants) | 292 | 284 | 242
  Month 12 | -1.4 (29.60) | -0.4 (31.64) | -2.6 (31.96)
  Month 18: number analyzed (Participants) | 236 | 227 | 174
  Month 18 | -2.3 (28.09) | -0.3 (31.04) | -1.1 (33.60)
  Discontinuation Visit: number analyzed (Participants) | 197 | 253 | 250
  Discontinuation Visit | -5.6 (34.29) | 1.8 (30.66) | -5.6 (33.73)

38. Secondary Outcome: Change From Baseline in the European Quality of Life-5 Dimensions (EQ-5D) Health Utility Index Score
Description: EQ-5D is a self-administered questionnaire that assesses health-related quality of life. The EQ-5D descriptive health profile comprises five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 3 levels of response: No problem (1), some problems (2), and extreme problems (3). A unique EQ-5D health state is defined by combining one level from each of the five dimensions into a single utility index score. EQ-5D index values range from -0.59 to 1.00 where higher EQ-5D scores represent better health status. A positive change from baseline score indicates improvement in health status and better health state.
Time Frame: Cycle 1 Day 1 (Baseline), then Months 1, 3, 6, 12, 18 and Discontinuation visit
Population: ITT population with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 490 | 492 | 490
units on a scale
  Month 1: number analyzed (Participants) | 400 | 420 | 381
  Month 1 | 0.0 (0.29) | -0.0 (0.31) | 0.0 (0.28)
  Month 3: number analyzed (Participants) | 389 | 283 | 366
  Month 3 | 0.1 (0.33) | 0.1 (0.32) | 0.1 (0.32)
  Month 6: number analyzed (Participants) | 341 | 351 | 323
  Month 6 | 0.1 (0.32) | 0.1 (0.31) | 0.1 (0.34)
  Month 12: number analyzed (Participants) | 283 | 278 | 231
  Month 12 | 0.1 (0.33) | 0.1 (0.31) | 0.1 (0.35)
  Month 18: number analyzed (Participants) | 219 | 230 | 170
  Month 18 | 0.1 (0.36) | 0.1 (0.32) | 0.1 (0.35)
  Discontinuation Visit: number analyzed (Participants) | 186 | 231 | 240
  Discontinuation Visit | 0.0 (0.40) | 0.0 (0.35) | 0.0 (0.39)

39. Secondary Outcome: Healthcare Resource Utilization (HRU): Rate of Inpatient Hospitalizations Per Year
Description: HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU Analysis may help in evaluating potential costs and budget impact of new treatments from a payer perspective. The rate of inpatient hospitalizations per patient year was calculated as the total number of hospitalizations divided by the total number of patient-years followed in the study period. Patient-years (PY) were calculated as the duration from baseline to last available HRQL assessment for each patient.
Time Frame: Day 1 (randomization) up to last visit completed 25 July 2016
Population: Healthcare Resource Utilization not analyzed.
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Number of Participants With Adverse Events (AEs) During the Active Treatment Phase
Description: A TEAE is any AE occurring or worsening on or after the first treatment of any study drug, and within 30 days after the last dose of the last study drug. Severity grades according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) on a 1-5 scale: Grade 1= Mild AE, Grade 2= Moderate AE, Grade 3= Severe AE, Grade 4= Life-threatening or disabling AE, Grade 5=Death related to AE. A serious AE is any AE occurring at any dose that: • Results in death; • Is life-threatening; • Requires or prolongs existing inpatient hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Constitutes an important medical event.
Time Frame: From first dose of study drug through 28 days following the discontinuation visit from active treatment phase; median duration of treatment was 80.2 weeks in the Rd arm; 72 weeks in the Rd18 arm and 67.1 weeks in the MPT arm
Population: Safety population included all participants who received at least one dose treatment dose of treatment in any arm
Measure: Number; unit: Participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 532 | 540 | 541
Participants
  ≥ 1 adverse event (AE) | 529 | 536 | 539
  ≥ 1 grade (Gr) 3 or 4 AE | 453 | 433 | 480
  ≥ 1 grade (Gr) 5 AE | 50 | 36 | 38
  ≥ 1 serious adverse event (SAE) | 359 | 308 | 270
  ≥ 1 AE related to Lenalidomide/Dex/Mel/Pred/Thal | 506 | 501 | 527
  ≥ 1 AE related to Lenalidomide | 482 | 481 | 0
  ≥ 1 AE related to dexamethasone | 429 | 410 | 0
  ≥ 1 AE related to melphalan | 0 | 0 | 441
  ≥ 1 AE related to prednisone | 0 | 0 | 326
  ≥ 1 AE related to thalidomide | 0 | 0 | 493
  ≥1 AE related to Lenalidomide/Dex or Mel/Pred/Thal | 269 | 269 | 145
  ≥ 1 Gr 3 or 4 AE related to Len/Dex/Mel/Pred/Thal | 373 | 326 | 423
  ≥ 1 grade 3 or 4 AE related to Lenalidomide | 342 | 290 | 0
  ≥ 1 grade 3 or 4 AE related to dexamethasone | 229 | 177 | 0
  ≥ 1 grade 3 or 4 AE related to melphalan | 0 | 0 | 307
  ≥ 1 grade 3 or 4 AE related to prednisone | 0 | 0 | 118
  ≥ 1 grade 3 or 4 AE related to Thalidomide | 0 | 0 | 316
  ≥1Gr 3 or 4 AE related to Len/Dex or Mel/Pred/Thal | 131 | 104 | 49
  ≥ 1 Grade 5 AE related to Len/Dex/Mel/Pred/Thal | 17 | 11 | 10
  ≥ 1 Grade 5 AE related to Lenalidomide | 12 | 9 | 0
  ≥ 1 Grade 5 AE related to Dexamethasone | 16 | 7 | 0
  ≥ 1 Grade 5 AE related to melphalan | 0 | 0 | 6
  ≥ 1 Grade 5 AE related to prednisone | 0 | 0 | 5
  ≥ 1 Grade 5 AE related to Thalidomide | 0 | 0 | 5
  ≥1 Grade 5 AE related to Len/Dex or Mel/Pred/Thal | 11 | 5 | 2
  ≥1 SAE related to Len/Dex/Mel/Pred/Thal | 195 | 158 | 142
  ≥1 SAE related to Lenalidomide | 165 | 130 | 0
  ≥1 SAE related to dexamethasone | 130 | 97 | 0
  ≥1 SAE related to melphalan | 0 | 0 | 75
  ≥1 SAE related to prednisone | 0 | 0 | 62
  ≥1 SAE related to thalidomide | 0 | 0 | 94
  ≥1 SAE related to Len/Dex or Mel/Pred/Thal | 95 | 64 | 27
  ≥1AE leading to Len/Dex/Mel/Pred/Thal Withdrawal | 157 | 109 | 153
  ≥1 AE leading to Lenalidomide withdrawal | 109 | 93 | 0
  ≥1 AE leading to dexamethasone withdrawal | 152 | 104 | 0
  ≥1 AE leading to melphalan withdrawal | 0 | 0 | 83
  ≥1 AE leading to prednisone withdrawal | 0 | 0 | 78
  ≥1 AE leading to Thalidomide withdrawal | 0 | 0 | 146
  ≥1AE leading to Len/DexOR Mel/Pred/Thal Withdrawal | 96 | 84 | 71
  ≥1AE leading to Len/Dex/Mel/Pred/Thal reduction | 279 | 214 | 348
  ≥1 AE leading to Lenalidomide reduction | 203 | 155 | 0
  ≥1 AE leading to dexamethasone reduction | 170 | 118 | 0
  ≥1 AE leading to melphalan reduction | 0 | 0 | 199
  ≥1 AE leading to prednisone reduction | 0 | 0 | 47
  ≥1 AE leading to thalidomide reduction | 0 | 0 | 254
  ≥1AE leading to Len/Dex or Mel/Pred/Thal reduction | 30 | 20 | 2
  ≥1 AE leading to Rd or MPT interruption | 368 | 321 | 419
  ≥1 AE leading to Lenalidomide interruption | 353 | 301 | 0
  ≥1 AE leading to dexamethasone interruption | 319 | 280 | 0
  ≥1 AE leading to melphalan interruption | 0 | 0 | 328
  ≥1 AE leading to prednisone interruption | 0 | 0 | 324
  ≥1 AE leading to Thalidomide interruption | 0 | 0 | 388
  ≥1 AE leading to Len and Dex or MPT interruption | 290 | 241 | 249

41. Secondary Outcome: Shift From Baseline to Most Extreme Postbaseline Value in Creatinine Clearance (CrCl) During the Active Treatment Phase
Description: Renal function was assessed for participants from baseline to the most extreme value in creatinine clearance calculated using the Cockcroft-Gault estimation.
Time Frame: Randomization to end of treatment or the data cut off of 24 May 2013; median duration of treatment was 80.2 weeks in the Rd arm; 72 weeks in the Rd18 arm and 67.1 weeks in the MPT arm
Population: Safety Population with baseline and postbaseline CrCl data.
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 494 | 506 | 484
participants
  CrCl< 30 mL/min to CrCl< 30 mL/min | 15 | 17 | 19
  CrCl < 30 mL/min to CrCl ≥ 30 but < 50 mL/min | 18 | 14 | 19
  CrCl < 30 mL/min to CrCl ≥ 50 but < 80 mL/min | 7 | 8 | 5
  CrCl< 30 mL/min to ≥ 80 mL/min | 2 | 2 | 0
  CrCl≥ 30 but < 50 mL/min to < 30 mL/min | 1 | 2 | 0
  CrCl ≥ 30 but < 50 mL/min to CrCl ≥ 30 but < 50 mL | 37 | 41 | 41
  CrCl ≥ 30 but < 50 mL/min to CrCl ≥ 50 but < 80 mL | 67 | 55 | 65
  CrCl ≥ 30 but < 50 mL/min to ≥ 80 mL/min | 9 | 12 | 2
  CrCl ≥ 50 but < 80 mL to CrCl< 30 mL/min | 0 | 0 | 0
  CrCl ≥ 50 but < 80 mL to CrCl ≥ 30 but < 50 mL/min | 4 | 1 | 4
  CrCl ≥ 50 but < 80 mL to CrCl ≥ 50 but < 80 mL/min | 112 | 130 | 102
  CrCl ≥ 50 but < 80 mL to ≥ 80 mL/min | 107 | 99 | 97
  CrCl ≥ 80 mL/min to CrCl< 30 mL/min | 0 | 1 | 0
  CrCl ≥ 80 mL/min to CrCl ≥ 30 but < 50 mL/min | 0 | 0 | 0
  CrCl ≥ 80 mL/min to CrCl ≥ 50 but < 80 mL/min | 6 | 10 | 9
  CrCl ≥ 80 mL/min to CrCl ≥ 80 mL/min | 109 | 114 | 121

42. Secondary Outcome: Shift From Baseline to Most Extreme Postbaseline Value in Absolute Neutrophil Count During the Active Treatment Phase
Description: Neutrophil counts was assessed for participants from baseline grade to most extreme severity grade using the NCI CTCAE v 3.0 grading scale.
Time Frame: as for outcome 41
Population: Safety Population; includes participants with baseline and postbaseline absolute neutrophil laboratory test grade information
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 525 | 534 | 526
participants
  Normal Baseline Grade to Normal Postbaseline Grade | 103 | 133 | 37
  Normal Baseline Grade to Grade 1 postbaseline | 96 | 85 | 79
  Normal Baseline Grade to Grade 2 postbaseline | 121 | 109 | 128
  Normal Baseline Grade to Grade 3 postbaseline | 70 | 71 | 141
  Normal Baseline Grade to Grade 4 postbaseline | 21 | 30 | 45
  Grade 1 Baseline to Normal postbaseline | 7 | 6 | 2
  Grade1 Baseline to Grade 1 postbaseline | 8 | 11 | 2
  Grade 1 Baseline to Grade 2 postbaseline | 17 | 15 | 11
  Grade 1 Baseline to Grade 3 postbaseline | 25 | 30 | 20
  Grade 1 Baseline to Grade 4 postbaseline | 9 | 4 | 21
  Grade 2 Baseline to normal postbaseline | 1 | 0 | 0
  Grade 2 Baseline to Grade 1 postbaseline | 1 | 1 | 1
  Grade 2 Baseline to Grade 2 postbaseline | 14 | 11 | 7
  Grade 2 Baseline to Grade 3 postbaseline | 18 | 18 | 21
  Grade 2 Baseline to Grade 4 postbaseline | 9 | 5 | 10
  Grade 3 Baseline to Normal postbaseline | 0 | 0 | 0
  Grade 3 Baseline to Grade 1 postbaseline | 0 | 0 | 0
  Grade 3 Baseline to Grade 2 postbaseline | 2 | 1 | 0
  Grade 3 Baseline to Grade 3 postbaseline | 2 | 2 | 0
  Grade3 Baseline to Grade 4 postbaseline | 0 | 2 | 1
  Grade 4 Baseline to Normal postbaseline Grade | 0 | 0 | 0
  Grade 4 Baseline to Grade 1 postbaseline Grade | 1 | 0 | 0
  Grade 4 Baseline to Grade 2 postbaseline | 0 | 0 | 0
  Grade 4 Baseline Grade to Grade 3 postbaseline | 0 | 0 | 0
  Grade 4 Baseline to Grade 4 postbaseline | 0 | 0 | 0

43. Secondary Outcome: Shift From Baseline to Most Extreme Postbaseline Value in Hemoglobin During the Active Treatment Phase
Description: Hemoglobin was assessed for participants from baseline grade to most extreme severity grade using the NCI CTCAE v 3.0 grading scale.
Time Frame: as for outcome 41
Population: Safety Population; Includes participants with baseline and postbaseline hemoglobin laboratory test grade information
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 527 | 535 | 526
participants
  Normal Baseline Grade to Normal Postbaseline Grade | 6 | 10 | 9
  Normal Baseline Grade to Grade 1 postbaseline | 39 | 30 | 25
  Normal Baseline Grade to Grade 2 postbaseline | 8 | 8 | 4
  Normal Baseline Grade to Grade 3 postbaseline | 0 | 1 | 1
  Normal Baseline Grade to Grade 4 postbaseline | 0 | 0 | 0
  Grade 1 Baseline to Normal postbaseline | 0 | 0 | 0
  Grade 1 Baseline to Grade 1 postbaseline | 106 | 126 | 110
  Grade1 Baseline to Grade 2 postbaseline | 128 | 123 | 123
  Grade 1 Baseline to Grade 3 postbaseline | 25 | 17 | 20
  Grade 1 Baseline to Grade 4 postbaseline | 2 | 5 | 4
  Grade 2 Baseline to normal postbaseline | 0 | 0 | 0
  Grade 2 Baseline to Grade 1 postbaseline | 8 | 12 | 14
  Grade 2 Baseline to Grade 2 postbaseline | 125 | 135 | 133
  Grade 2 Baseline to Grade 3 postbaseline | 48 | 41 | 47
  Grade 2 Baseline to Grade 4 postbaseline | 4 | 9 | 11
  Grade 3 Baseline to Normal postbaseline | 0 | 0 | 0
  Grade 3 Baseline to Grade 1 postbaseline | 0 | 1 | 0
  Grade 3 Baseline to Grade 2 postbaseline | 12 | 4 | 10
  Grade 3 Baseline to Grade 3 postbaseline | 10 | 8 | 10
  Grade 3 Baseline to Grade 4 postbaseline | 5 | 3 | 2
  Grade 4 Baseline to Normal postbaseline | 0 | 0 | 0
  Grade 4 Baseline to Grade 1 postbaseline | 0 | 0 | 0
  Grade 4 Baseline to Grade 2 postbaseline | 0 | 0 | 1
  Grade 4 Baseline to Grade 3 postbaseline | 0 | 1 | 0
  Grade 4 Baseline to Grade 4 postbaseline | 1 | 1 | 2

44. Secondary Outcome: Shift From Baseline to Most Extreme Postbaseline Value in Platelet Count During the Active Treatment Phase.
Description: Improvement in platelets was assessed for participants from baseline grade to most extreme severity grade using the NCI CTCAE v 3.0 grading scale.
Time Frame: as for outcome 41
Population: Safety population; Includes participants with baseline and postbaseline platelet laboratory test grade information
Measure: Number; unit: participants
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 527 | 535 | 526
participants
  Normal Baseline Grade to Normal Postbaseline Grade | 197 | 197 | 165
  Normal Baseline Grade to Grade 1 postbaseline | 216 | 211 | 208
  Normal Baseline Grade to Grade 2 postbaseline | 24 | 30 | 27
  Normal Baseline Grade to Grade 3 postbaseline | 15 | 12 | 31
  Normal Baseline Grade to Grade 4 postbaseline | 4 | 5 | 11
  Grade1 Baseline to Normal postbaseline Grade | 1 | 3 | 6
  Grade 1 Baseline to Grade 1 postbaseline | 34 | 38 | 51
  Grade 1 Baseline to Grade 2 postbaseline | 15 | 19 | 7
  Grade 1 Baseline to Grade 3 postbaseline | 10 | 12 | 10
  Grade 1 Baseline to Grade 4 postbaseline | 2 | 1 | 1
  Grade 2 Baseline to normal postbaseline Grade | 0 | 0 | 0
  Grade 2 Baseline to Grade 1 postbaseline | 0 | 1 | 2
  Grade 2 Baseline to Grade 2 postbaseline | 3 | 3 | 1
  Grade 2 Baseline to Grade 3 postbaseline | 3 | 2 | 2
  Grade 2 Baseline to Grade 4 postbaseline | 1 | 0 | 2
  Grade 3 Baseline to Normal postbaseline Grade | 0 | 0 | 0
  Grade 3 Baseline to Grade 1 postbaseline | 0 | 0 | 0
  Grade 3 Baseline to Grade 2 postbaseline | 0 | 0 | 1
  Grade 3 Baseline to Grade 3 postbaseline | 0 | 0 | 1
  Grade 3 Baseline to Grade 4 postbaseline | 2 | 1 | 0

45. Secondary Outcome: Improvement of Infection Rate by Observing the Historical Data Compared to the Clinical Data Base
Description: Improvement of infection rate by observing historical data compared to the data within clinical database as not analyzed.
Time Frame: From randomization to 24 May 2013
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone Rd18 | Melphalan + Prednisone + Thalidomide (MPT)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of treatment to at least 28 days after discontinuation of active treatment for those not continuing in the PFS phase; median duration of treatment was 80.2 weeks in the Rd arm, 72.0 weeks in the Rd18 arm and 67.1 weeks in the MPT arm.
Groups:
- Lenalidomide and Dexamethasone (Rd18): Participants ≤ 75 years old received 25 mg lenalidomide (R) PO on days 1 to 21 of each 28-day treatment cycle 40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless progressive disease (PD) or intolerable toxicity occurred. Those > 75 years old received lenalidomide 25 mg PO on the same schedule and frequency plus 20 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity. Those with moderate renal insufficiency received 10-15 mg lenalidomide (R) PO on days 1-21 of each 28-day cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity. Participants with severe renal insufficiency received 15 mg lenalidomide (R) PO every other day (QOD) on days 1-21 of each 28-day cycle and 20-40 mg dexamethasone (d) PO on days 1, 8, 15, and 22 of a 28-day cycle for up to 18 cycles unless PD or intolerable toxicity.
Arm/Group | Lenalidomide and Low-Dose Dexamethasone (Rd) | Lenalidomide and Dexamethasone (Rd18) | Melphalan + Prednisone + Thalidomide (MPT)
Serious Adverse Events (participants affected / at risk) | 378/532 | 308/540 | 270/541
Other Adverse Events (participants affected / at risk) | 523/532 | 532/540 | 532/541
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Low-Dose Dexamethasone (Rd) (N=532) | Lenalidomide and Dexamethasone (Rd18) (N=540) | Melphalan + Prednisone + Thalidomide (MPT) (N=541)
ANAEMIA (Blood and lymphatic system disorders) | 24 | 15 | 23
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 0 | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 2 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 8 | 13
HAEMOLYSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
HYPERVISCOSITY SYNDROME (Blood and lymphatic system disorders) | 1 | 0 | 0
HYPOCOAGULABLE STATE (Blood and lymphatic system disorders) | 0 | 0 | 1
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 3 | 4
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 1 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 5 | 7
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 | 6 | 10
ACUTE CORONARY SYNDROME (Cardiac disorders) | 5 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 6 | 1 | 4
ANGINA PECTORIS (Cardiac disorders) | 7 | 2 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 1
ARRHYTHMIA (Cardiac disorders) | 0 | 2 | 2
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 1 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 18 | 12 | 9
ATRIAL FLUTTER (Cardiac disorders) | 3 | 2 | 2
ATRIAL THROMBOSIS (Cardiac disorders) | 0 | 1 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 0 | 1
BRADYARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 2 | 2 | 2
CARDIAC AMYLOIDOSIS (Cardiac disorders) | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 5 | 3 | 1
CARDIAC FAILURE (Cardiac disorders) | 13 | 11 | 8
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 7 | 5 | 5
CARDIAC FLUTTER (Cardiac disorders) | 0 | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 2 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 2 | 1 | 1
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 2
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0
COR PULMONALE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 5 | 0 | 0
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 1 | 2
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 0 | 1 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 2 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 7 | 2 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 0 | 0
NODAL ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
PERICARDITIS (Cardiac disorders) | 0 | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 1 | 0 | 0
SINOATRIAL BLOCK (Cardiac disorders) | 0 | 0 | 1
SINUS ARREST (Cardiac disorders) | 1 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 2 | 0 | 2
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 2 | 2
TACHYARRHYTHMIA (Cardiac disorders) | 2 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 4 | 0
VENTRICULAR FLUTTER (Cardiac disorders) | 0 | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
LEFT VENTRICLE OUTFLOW TRACT OBSTRUCTION (Congenital, familial and genetic disorders) | 0 | 0 | 1
THALASSAEMIA BETA (Congenital, familial and genetic disorders) | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 1 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0
THYROID CYST (Endocrine disorders) | 0 | 0 | 1
BLINDNESS UNILATERAL (Eye disorders) | 1 | 0 | 0
CATARACT (Eye disorders) | 5 | 0 | 1
CHOROIDAL DETACHMENT (Eye disorders) | 0 | 1 | 0
CONJUNCTIVAL OEDEMA (Eye disorders) | 0 | 1 | 0
DIABETIC RETINOPATHY (Eye disorders) | 1 | 0 | 0
DIPLOPIA (Eye disorders) | 1 | 1 | 0
GLAUCOMA (Eye disorders) | 0 | 1 | 0
OCULAR HYPERTENSION (Eye disorders) | 0 | 1 | 0
UVEITIS (Eye disorders) | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 1 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 1 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 | 0
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2 | 0 | 0
COLONIC POLYP (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 5 | 3 | 5
DIARRHOEA (Gastrointestinal disorders) | 9 | 8 | 4
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 2 | 1 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
ENTERITIS (Gastrointestinal disorders) | 0 | 1 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 0 | 0 | 1
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0 | 0
FAECALOMA (Gastrointestinal disorders) | 0 | 3 | 0
GASTRIC DISORDER (Gastrointestinal disorders) | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 3 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 0 | 0
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 2 | 0 | 0
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 1 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1 | 0
HAEMORRHAGIC EROSIVE GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
ILEUS (Gastrointestinal disorders) | 0 | 0 | 3
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 3 | 2 | 1
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 1 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 4 | 3 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 2 | 7
NECROTISING COLITIS (Gastrointestinal disorders) | 1 | 0 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 | 0 | 0
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1 | 1
ORAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 1 | 0
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0
RECTAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
REFLUX GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
SIGMOIDITIS (Gastrointestinal disorders) | 1 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1 | 2
SUBILEUS (Gastrointestinal disorders) | 0 | 1 | 0
TONGUE HAEMATOMA (Gastrointestinal disorders) | 0 | 1 | 0
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1
VOMITING (Gastrointestinal disorders) | 8 | 4 | 8
ASTHENIA (General disorders) | 12 | 2 | 5
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 0 | 1
CHILLS (General disorders) | 1 | 1 | 0
DEATH (General disorders) | 3 | 3 | 1
FATIGUE (General disorders) | 3 | 3 | 3
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 16 | 13 | 12
GENERALISED OEDEMA (General disorders) | 1 | 1 | 0
HYPERPYREXIA (General disorders) | 0 | 1 | 0
HYPERTHERMIA (General disorders) | 0 | 1 | 0
HYPOTHERMIA (General disorders) | 0 | 0 | 1
INFLAMMATION (General disorders) | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0
INJECTION SITE HAEMORRHAGE (General disorders) | 1 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 2
MUCOSAL INFLAMMATION (General disorders) | 1 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 3 | 3
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 4 | 1
OEDEMA PERIPHERAL (General disorders) | 5 | 2 | 3
PAIN (General disorders) | 5 | 0 | 4
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 1 | 1
PYREXIA (General disorders) | 22 | 11 | 8
SPINAL PAIN (General disorders) | 0 | 1 | 1
SUDDEN DEATH (General disorders) | 5 | 2 | 2
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0 | 0
ULCER HAEMORRHAGE (General disorders) | 0 | 0 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 1 | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 0
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0 | 0
AMYLOIDOSIS (Immune system disorders) | 1 | 0 | 0
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 1 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0 | 0
ANORECTAL INFECTION BACTERIAL (Infections and infestations) | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 1
ARTHRITIS BACTERIAL (Infections and infestations) | 5 | 0 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 1 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 1 | 0
BACTERAEMIA (Infections and infestations) | 3 | 2 | 2
BACTERIAL SEPSIS (Infections and infestations) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 13 | 6 | 2
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 5 | 2
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 | 1 | 0
BURSITIS INFECTIVE STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0
CAMPYLOBACTER INFECTION (Infections and infestations) | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 8 | 3 | 2
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 1 | 0 | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 2 | 0 | 2
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 2 | 1 | 1
DOUGLAS' ABSCESS (Infections and infestations) | 0 | 1 | 0
EMBOLIC PNEUMONIA (Infections and infestations) | 1 | 0 | 0
ENDOCARDITIS (Infections and infestations) | 0 | 0 | 1
ENDOCARDITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
ENDOCARDITIS STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 0
ENDOPHTHALMITIS (Infections and infestations) | 0 | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 3 | 1 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 3 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0
FUNGAL INFECTION (Infections and infestations) | 1 | 1 | 0
FURUNCLE (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 3 | 2
GASTROENTERITIS SALMONELLA (Infections and infestations) | 1 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 2
HERPES ZOSTER (Infections and infestations) | 3 | 1 | 1
INFECTION (Infections and infestations) | 4 | 1 | 4
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 4 | 0 | 0
INFECTIVE TENOSYNOVITIS (Infections and infestations) | 0 | 1 | 0
INFLUENZA (Infections and infestations) | 7 | 3 | 1
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 | 0 | 0
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 1 | 0 | 0
KLEBSIELLA INFECTION (Infections and infestations) | 0 | 0 | 1
KLEBSIELLA SEPSIS (Infections and infestations) | 0 | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 8 | 7 | 3
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 3 | 4
LUNG INFECTION (Infections and infestations) | 3 | 8 | 5
LUNG INFECTION PSEUDOMONAL (Infections and infestations) | 0 | 0 | 2
MENINGITIS (Infections and infestations) | 0 | 1 | 0
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 1 | 0 | 0
MENINGOCOCCAL SEPSIS (Infections and infestations) | 1 | 0 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 2 | 1 | 2
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 | 1 | 0
ORCHITIS (Infections and infestations) | 1 | 1 | 0
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0
PERIODONTITIS (Infections and infestations) | 1 | 0 | 0
PERIORBITAL ABSCESS (Infections and infestations) | 1 | 0 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 1 | 0 | 0
PERITONITIS (Infections and infestations) | 1 | 1 | 0
PNEUMOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 3 | 0 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 3 | 0 | 1
PNEUMONIA (Infections and infestations) | 60 | 48 | 35
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 2
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 | 1 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 1 | 0 | 0
PNEUMONIA LEGIONELLA (Infections and infestations) | 2 | 1 | 1
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 4 | 2 | 1
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 2 | 0 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 1 | 0
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 1
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 | 0 | 0
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 | 0 | 0
PROSTATIC ABSCESS (Infections and infestations) | 0 | 1 | 0
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 1 | 0 | 0
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 1 | 1
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 4 | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 5 | 4
SEPSIS (Infections and infestations) | 17 | 10 | 8
SEPTIC SHOCK (Infections and infestations) | 5 | 7 | 3
SINUSITIS (Infections and infestations) | 1 | 0 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 0 | 1 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 4 | 0 | 0
STAPHYLOCOCCAL IMPETIGO (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 | 3 | 0
STRONGYLOIDIASIS (Infections and infestations) | 1 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 | 0 | 0
TOOTH ABSCESS (Infections and infestations) | 0 | 1 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 1 | 0 | 0
TUBERCULOSIS (Infections and infestations) | 1 | 0 | 0
TUBERCULOUS PLEURISY (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 9 | 2
URINARY TRACT INFECTION (Infections and infestations) | 9 | 5 | 3
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1
UROSEPSIS (Infections and infestations) | 3 | 1 | 0
WHIPPLE'S DISEASE (Infections and infestations) | 1 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 | 1 | 2
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 | 1 | 0
BLADDER INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 2
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
FACE INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1
FALL (Injury, poisoning and procedural complications) | 5 | 3 | 4
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 3 | 2 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 6 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 2 | 1 | 0
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 0 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
HEART INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 4 | 2 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 6 | 1 | 1
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 1 | 0
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 2
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 | 0 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
RESPIRATORY FUME INHALATION DISORDER (Injury, poisoning and procedural complications) | 1 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 2 | 3 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 6 | 3 | 5
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 2
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 2
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 0
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
TRAUMATIC FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 2
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
BIOPSY BONE MARROW ABNORMAL (Investigations) | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 2 | 2 | 0
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 1 | 0 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
HAEMOGLOBIN ABNORMAL (Investigations) | 1 | 0 | 0
HEART RATE INCREASED (Investigations) | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 0
PROTEIN URINE PRESENT (Investigations) | 1 | 0 | 0
PROTHROMBIN TIME RATIO INCREASED (Investigations) | 0 | 1 | 0
TROPONIN INCREASED (Investigations) | 1 | 0 | 0
TROPONIN T INCREASED (Investigations) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 3 | 1 | 1
CACHEXIA (Metabolism and nutrition disorders) | 2 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 7 | 9 | 7
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 | 2 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1 | 1
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0 | 0
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 0 | 0 | 1
GOUT (Metabolism and nutrition disorders) | 3 | 1 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 5 | 10 | 7
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 3 | 0
HYPERGLYCAEMIC HYPEROSMOLAR NONKETOTIC SYNDROME (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 2 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 5 | 4 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 | 1 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 6 | 6 | 1
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0
MARASMUS (Metabolism and nutrition disorders) | 1 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 1
METABOLIC ALKALOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0
SHOCK HYPOGLYCAEMIC (Metabolism and nutrition disorders) | 1 | 0 | 0
TETANY (Metabolism and nutrition disorders) | 1 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 22 | 19 | 10
BONE LESION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 10 | 6 | 6
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
GOUTY TOPHUS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SOFT TISSUE MASS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
VERTEBRAL WEDGING (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 4 | 1
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
BOWEN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CARCINOID TUMOUR OF THE APPENDIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
COLON CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
ENDOMETRIAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
ENDOMETRIAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
GASTROINTESTINAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
LEUKAEMIA PLASMACYTIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG ADENOCARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
LUNG SQUAMOUS CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
NEOPLASM SWELLING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
ORAL NEOPLASM BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SMALL INTESTINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 5 | 1
TRANSITIONAL CELL CANCER OF THE RENAL PELVIS AND URETER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 2 | 0
BRAIN STEM INFARCTION (Nervous system disorders) | 1 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 0 | 0
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 1 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 4 | 1 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 2 | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 8 | 3 | 3
COMA (Nervous system disorders) | 0 | 1 | 0
CONVULSION (Nervous system disorders) | 3 | 0 | 0
COORDINATION ABNORMAL (Nervous system disorders) | 0 | 0 | 1
DEMENTIA (Nervous system disorders) | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 5 | 0 | 3
DYSTONIA (Nervous system disorders) | 1 | 0 | 1
EPIDURITIS (Nervous system disorders) | 1 | 1 | 0
EPILEPSY (Nervous system disorders) | 2 | 1 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 1 | 0
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 | 0 | 0
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 1
HEMIPARESIS (Nervous system disorders) | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 1 | 1
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 4 | 0 | 0
LACUNAR INFARCTION (Nervous system disorders) | 1 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 2 | 1
MOTOR NEURONE DISEASE (Nervous system disorders) | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1
PARALYSIS (Nervous system disorders) | 0 | 0 | 1
PARAPARESIS (Nervous system disorders) | 0 | 2 | 0
PARAPLEGIA (Nervous system disorders) | 0 | 1 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 1
PARKINSONISM (Nervous system disorders) | 0 | 1 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 1 | 0 | 0
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 | 1 | 0
PRESYNCOPE (Nervous system disorders) | 6 | 1 | 2
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 | 1 | 0
RADICULITIS (Nervous system disorders) | 1 | 0 | 0
REPETITIVE SPEECH (Nervous system disorders) | 1 | 0 | 0
SCIATICA (Nervous system disorders) | 1 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0
SPEECH DISORDER (Nervous system disorders) | 1 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 9 | 3 | 8
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 0 | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 | 2 | 2
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 | 0 | 1
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 1 | 0 | 0
AGITATED DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 2
COMPLETED SUICIDE (Psychiatric disorders) | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 7 | 6 | 2
DELIRIUM (Psychiatric disorders) | 4 | 2 | 1
DEPRESSED MOOD (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 4 | 2 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 2 | 0
EUPHORIC MOOD (Psychiatric disorders) | 1 | 0 | 0
HALLUCINATION (Psychiatric disorders) | 0 | 1 | 0
IMPAIRED SELF-CARE (Psychiatric disorders) | 0 | 1 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 | 1 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
AZOTAEMIA (Renal and urinary disorders) | 1 | 1 | 0
BLADDER PROLAPSE (Renal and urinary disorders) | 1 | 0 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 1
OLIGURIA (Renal and urinary disorders) | 1 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 1
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 | 1 | 0
RENAL COLIC (Renal and urinary disorders) | 2 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 8 | 18 | 14
RENAL FAILURE ACUTE (Renal and urinary disorders) | 21 | 16 | 10
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 1 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 5 | 2 | 4
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 2 | 4 | 2
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 | 1 | 0
GENITAL PROLAPSE (Reproductive system and breast disorders) | 0 | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 1 | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 8
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 20 | 15 | 20
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY ALKALOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 4
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
ACUTE FEBRILE NEUTROPHILIC DERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
CUTANEOUS VASCULITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRUG RASH WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 5 | 5 | 3
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 1 | 0 | 0
AORTIC DISSECTION (Vascular disorders) | 1 | 0 | 0
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 19 | 11 | 8
HAEMATOMA (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 2
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0 | 1
HYPOTENSION (Vascular disorders) | 8 | 7 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 3 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 | 1 | 0
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 | 0 | 1
PHLEBITIS (Vascular disorders) | 2 | 0 | 5
SHOCK (Vascular disorders) | 1 | 0 | 0
THROMBOPHLEBITIS (Vascular disorders) | 1 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide and Low-Dose Dexamethasone (Rd) (N=532) | Lenalidomide and Dexamethasone (Rd18) (N=540) | Melphalan + Prednisone + Thalidomide (MPT) (N=541)
ANAEMIA (Blood and lymphatic system disorders) | 237 | 191 | 219
LEUKOPENIA (Blood and lymphatic system disorders) | 66 | 59 | 92
LYMPHOPENIA (Blood and lymphatic system disorders) | 60 | 43 | 71
NEUTROPENIA (Blood and lymphatic system disorders) | 194 | 177 | 325
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 111 | 99 | 132
ATRIAL FIBRILLATION (Cardiac disorders) | 30 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 27 | 0 | 35
CATARACT (Eye disorders) | 84 | 31 | 0
VISION BLURRED (Eye disorders) | 30 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 68 | 40 | 28
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 50 | 34 | 29
CONSTIPATION (Gastrointestinal disorders) | 233 | 210 | 282
DIARRHOEA (Gastrointestinal disorders) | 248 | 205 | 86
DRY MOUTH (Gastrointestinal disorders) | 38 | 38 | 62
DYSPEPSIA (Gastrointestinal disorders) | 59 | 28 | 36
NAUSEA (Gastrointestinal disorders) | 156 | 127 | 163
TOOTHACHE (Gastrointestinal disorders) | 28 | 0 | 0
VOMITING (Gastrointestinal disorders) | 97 | 66 | 104
ASTHENIA (General disorders) | 148 | 122 | 123
FATIGUE (General disorders) | 178 | 176 | 153
NON-CARDIAC CHEST PAIN (General disorders) | 31 | 27 | 0
OEDEMA (General disorders) | 38 | 28 | 32
OEDEMA PERIPHERAL (General disorders) | 220 | 168 | 213
PYREXIA (General disorders) | 111 | 94 | 69
BRONCHITIS (Infections and infestations) | 90 | 57 | 42
GASTROENTERITIS (Infections and infestations) | 35 | 0 | 0
INFLUENZA (Infections and infestations) | 33 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 29 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 90 | 54 | 33
PNEUMONIA (Infections and infestations) | 29 | 34 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 35 | 0 | 0
RHINITIS (Infections and infestations) | 31 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 71 | 48 | 31
URINARY TRACT INFECTION (Infections and infestations) | 77 | 59 | 38
CONTUSION (Injury, poisoning and procedural complications) | 39 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 46 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 39 | 0 | 0
WEIGHT DECREASED (Investigations) | 73 | 78 | 47
DECREASED APPETITE (Metabolism and nutrition disorders) | 128 | 115 | 72
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 61 | 50 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 60 | 54 | 30
HYPOKALAEMIA (Metabolism and nutrition disorders) | 104 | 62 | 38
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 27 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 110 | 71 | 67
BACK PAIN (Musculoskeletal and connective tissue disorders) | 175 | 137 | 115
BONE PAIN (Musculoskeletal and connective tissue disorders) | 83 | 72 | 58
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 29 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 115 | 102 | 61
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 46 | 34 | 28
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 63 | 51 | 39
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 72 | 58 | 36
MYALGIA (Musculoskeletal and connective tissue disorders) | 31 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 43 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 91 | 65 | 60
DIZZINESS (Nervous system disorders) | 87 | 70 | 114
DYSGEUSIA (Nervous system disorders) | 41 | 45 | 0
HEADACHE (Nervous system disorders) | 80 | 52 | 55
HYPOAESTHESIA (Nervous system disorders) | 46 | 0 | 40
NEUROPATHY PERIPHERAL (Nervous system disorders) | 35 | 0 | 62
PARAESTHESIA (Nervous system disorders) | 88 | 74 | 102
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 28 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 113 | 93 | 191
SOMNOLENCE (Nervous system disorders) | 31 | 0 | 51
TREMOR (Nervous system disorders) | 77 | 73 | 100
ANXIETY (Psychiatric disorders) | 45 | 36 | 41
CONFUSIONAL STATE (Psychiatric disorders) | 35 | 0 | 0
DEPRESSION (Psychiatric disorders) | 66 | 45 | 30
INSOMNIA (Psychiatric disorders) | 150 | 127 | 53
RENAL FAILURE (Renal and urinary disorders) | 27 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 129 | 94 | 67
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 31 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 112 | 85 | 110
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 30 | 28 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 32 | 31 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 32 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 35 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 32 | 30 | 36
ERYTHEMA (Skin and subcutaneous tissue disorders) | 35 | 27 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 49 | 49 | 0
RASH (Skin and subcutaneous tissue disorders) | 117 | 129 | 91
DEEP VEIN THROMBOSIS (Vascular disorders) | 40 | 0 | 0
HYPERTENSION (Vascular disorders) | 43 | 27 | 35
HYPOTENSION (Vascular disorders) | 52 | 28 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to ninety days; Investigator must delete confidential information before submission or defer publication to permit patent applications